#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | • | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for A Phase I, Randomized, Double-Blind (Sponsor Unblinded), Single-Center, Placebo-Controlled, Three-Part Study to Evaluate the Safety Tolerability, and Pharmacokinetics of Ascending Single and Repeat Intravenous Doses of GSK3342830 in Healthy Adul Subjects |
|---|---|---|
| <b>Compound Number</b> | : | GSK3342830 |
| Effective Date | · | 17-AUG-2017 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204847.
- This RAP is intended to describe the safety, tolerability, and pharmacokinetic analyses required for the study.
- This RAP is updated based upon Protocol Amendment 1. However,, Part 3 (Japanese subjects) that was added in Protocol Amendment 1 will not be conducted.
- This RAP will be provided to the study team members to convey the content of the Dose Escalation (DE) and Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD |
|---|
| Biostatistics Team Leader (Biostatistics, Early Development 28-AUG-2017 |
| Services) |
| PPD 29 ALIC 2017 |
| Senior Pharmacokineticist (Biostatistics) 28-AUG-2017 |

#### Approved by:

| PPD | | 28-AUG-2017 |
|-----------------|--------------------|-------------|
| Director Clinic | al Statistics, GSK | 26-AUG-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPO | PRTING & ANALYSIS PLAN SYNPOSIS | 4 |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | MARY OF KEY PROTOCOL INFORMATION | 7<br>7<br>9 |
| 3. | PLANN<br>3.1.<br>3.2. | NED ANALYSES<br>Interim Analyses<br>Final Analyses | 11 |
| 4. | ANALY<br>4.1. | YSIS POPULATIONSProtocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING /ENTIONS | 13 |
| 6. | STUD'<br>6.1. | Y POPULATION ANALYSES Overview of Planned Analyses | |
| 7. | PRIMA<br>7.1. | ARY STATISTICAL ANALYSESSafety Analyses7.1.1. Overview of Planned Safety Analyses | 15 |
| 8. | SECO<br>8.1. | Pharmacokinetic Analyses 8.1.1. Overview of Planned Pharmacokinetic Analyses 8.1.2. Drug Concentration Measures 8.1.3. Pharmacokinetic Parameters 8.1.3.1. Deriving Pharmacokinetic Parameters 8.1.3.2. Statistical Analysis of Pharmacokinetic Parameters | 17<br>17<br>17<br>17 |
| | 8.2. | Bayesian Dose Escalation Analyses | 22<br>22 |
| 9. | REFE | RENCES | 27 |
| 10. | APPEN<br>10.1. | 10.1.1. Protocol Defined Time & Events | 29<br>29 |
| | 10.2. | Appendix 2: Treatment States and Phases | 35<br>35<br>35 |
| | 10.3. | Appendix 3: Data Display Standards & Handling Conventions | |

## CONFIDENTIAL

| | 10.3.1. | Study Treat | ment & Sub-group Display Descriptors | 36 |
|---|---|---|---|---|
| | 10.3.2. | | finition & Derivations | |
| | | 10.3.2.1. E | Baseline Definitions | 37 |
| | | 10.3.2.2. [ | Derivations and Handling of Missing Baseline | |
| | | | Data | 37 |
| | 10.3.3. | Reporting P | rocess & Standards | 37 |
| 10.4. | Appendix | 4: Derived a | and Transformed Data | 40 |
| | 10.4.1. | General | | 40 |
| | 10.4.2. | Study Popul | ation | 40 |
| | 10.4.3. | Safety | | 40 |
| 10.5. | Appendix | 5: Prematur | e Withdrawals and Handling of Missing Data | 42 |
| | 10.5.1. | Premature V | Vithdrawals | 42 |
| | 10.5.2. | Handling of | Missing Data | 42 |
| | | 10.5.2.1. H | Handling of Missing Dates | 42 |
| | | | landling of Partial Dates | |
| 10.6. | <b>Appendix</b> | 6: Values of | f Potential Clinical Importance | 44 |
| | 10.6.1. | ECG | | 44 |
| | 10.6.2. | | | 44 |
| 10.7. | Appendix | 7: DMID Ad | ult Toxicity Tables for Adverse Event | |
| | Assessm | ent | | 45 |
| | | | /alues | |
| 10.8. | <b>Appendix</b> | 8: Multiple ( | Comparisons & Multiplicity | 48 |
| | 10.8.1. | | Multiple Comparisons & Multiplicity | 48 |
| 10.9. | <b>Appendix</b> | 9: Model Ch | necking and Diagnostics for Statistical | |
| | Analyses | | | |
| | 10.9.1. | | nalysis Assumptions | |
| 10.10. | | | viations & Trade Marks | |
| | | | ns | |
| 10.11. | | | ata Displays | |
| | | | y Numbering | |
| | | | ple Shell Referencing | |
| | | | [Priority] | |
| | | , , | ation Tables | |
| | | • | es | |
| | | | es | |
| | | | netic Tables | |
| | | | netic Figures | |
| | 10.11.9. | ICH Listings | S | 62 |

## 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe: |
| | <ul> <li>Any planned analyses and output to be included in the clinical study report for<br/>Protocol 204847.</li> </ul> |
| Protocol | This RAP is based on the original protocol (Dated: 18-FEB-2016) of study 204847 (GSK Document No. : 2015N257523_00). |
| Primary<br>Objective | For Part 1, to investigate the safety and tolerability of GSK3342830 after administration of single IV doses in healthy adult subjects |
| | For Part 2, to investigate the safety and tolerability of GSK3342830 after administration of repeat IV doses in healthy adult subjects |
| | For Part 3, to investigate the safety and tolerability of GSK3342830 after administration of a single IV dose in healthy adult Japanese subjects |
| Primary<br>Endpoint | Clinical safety data from adverse events (AEs), clinical laboratory tests, vital signs (blood pressure, heart rate, temperature, and respiration rate), and 12-lead electrocardiogram (ECG) readings |
| Study<br>Design | This is a Phase I, first-time-in-human (FTIH), randomized, double-blind (sponsor unblinded), single-center, placebo-controlled, dose-escalation study to determine the safety, tolerability, and pharmacokinetic (PK) profile of GSK3342830 after administration of single (Part 1) and repeat (Part 2) IV doses in healthy adult subjects, and after administration of a single IV dose in healthy adult Japanese subjects (Part 3). |
| | Dose escalation will be conducted only if it is supported by the preliminary safety, tolerability, and PK results from the preceding dose levels in the study. This is the first administration of GSK3342830 in humans; therefore, as preliminary safety, tolerability, and PK results are reviewed internally at GSK and with the clinical study site, study design adjustments may be made based on emerging data from each dose cohort. |
| | The repeat dose escalation component (Part 2) of this study is planned to be initiated after completion and evaluation of the all single dose cohorts up to and including 4000 mg. Initiation of Part 2 will be based on the evaluation of preliminary safety, tolerability, and PK data from the single dose escalation (Part 1) cohorts once safety at an exposure that exceeds the daily exposure predicted for the Part 2 planned starting dose of 1000 mg TID is demonstrated, which is predicted to occur at the 4000 mg single dose. |
| | The single dose administration in Japanese subjects component (Part 3) of this study is planned to be conducted in parallel with Part 2. The dose for the Part 3 cohort will be based on preliminary safety and tolerability results of doses determined to be safe and well tolerated in subjects of non-Japanese heritage after completion of the single escalation dose cohorts (Part 1). |
| Planned | Safety and PK data will be presented in tabular and/or graphical format and |

| Overview | Key Elements of the RAP |
|---|---|
| Analyses | summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. |
| Analysis<br>Populations | Safety Population – defined as all subjects who receive at least 1 dose of study drug and have at least 1 post-dose safety assessment. |
| | PK Population - defined as all subjects who receive at least 1 dose of GSK3342830 and have evaluable PK data for GSK3342830. |
| | PK Parameter Population - defined as all subjects in the PK population for whom valid and evaluable PK parameters were derived. |
| Hypothesis | No inferential hypothesis testing will be performed on the safety variables. |
| | <ul> <li>Dose proportionality of AUC(0-∞) and Cmax on Day 1 and for repeat dose<br/>groups AUC(0-τ) and Cmax of GSK3342830 on Day 15 will be assessed<br/>separately by day using the following power model:</li> </ul> |
| | y = a * doseβ. |
| | where y denotes the PK parameter being analyzed and a depends on the random error in the repeat dose phase where subjects take the study drug in a parallel-group fashion. Dose proportionality implies that $\beta$ =1 and will be assessed by estimating $\beta$ along with its 90% CI. The exponent, $\beta$ , in the power model will be estimated by regressing the loge-transformed PK parameter on loge-transformed dose. |
| | $log(y)=log(\alpha) + \beta * log(dose)$ |
| | The power model will be fitted by restricted maximum likelihood (REML) using Statistical Analysis Software (SAS) Proc Mixed, with a fixed effect term for dose. The PK parameter endpoint and the factor dose will be loge-transformed prior to the analysis. |
| | <ul> <li>For the repeat dose cohorts (Part 2), the time invariance ratio will be assessed by fitting a mixed effect model for AUC(0-∞) on Day 1 and AUC(0-τ) on Day 15 data with subject as a random effect and group (group=1 for AUC(0-∞) on Day 1, and group=2 for AUC(0-τ) on Day 15) as a fixed effect for each cohort.</li> </ul> |
| | For the repeat dose cohorts (Part 2), the accumulation ratio (Ro) will be calculated as the ratio of AUC(0-τ) on Day 15 to AUC(0-τ) on Day 1 for each subject. The dosing interval (τ) will be equal to 8 hours. Following log-transformation, AUC(0-τ) of GSK3342830 on Days 1 and 15 will be analyzed by a mixed effect model, fitting dose, day, and dose-by-day interaction as fixed effects and subject as a random effect. For each dose, point estimate and 90% CI for the difference "AUC(0-τ) on Day 15 - AUC(0-τ) on Day 1" will be constructed using the appropriate error term. The point estimate and associated 90% CI will then be exponentially back-transformed to provide point and 90% CI estimates for the ratios "AUC(0-τ) on Day 15: AUC(0-τ) on Day 1." If dose-by-day interaction is not significant, then a single point estimate and 90% CI pooled across all doses for the ratio AUC(0-τ) on Day 15: AUC(0-τ) on Day 1 |

| Overview | Key Elements of the RAP |
|---|---|
| | may be constructed with all estimates for each dose. |
| | • To evaluate whether steady state was achieved, statistical analysis of steady-state Cτ will be performed after log-transformation of Cτ on Days 3, 6, 9, 12, 13, and 15. A mixed effect model will be fitted by dose and day (as a continuous covariate) as a fixed effect term and subject as a random effect term. Distributional assumptions underlying the statistical analyses will be assessed by visual inspection of residual plots. Normality will be examined by normal probability plots, while homogeneity of variance will be assessed by plotting the residuals against the predicted values for the model. Alternative analyses of the data will be performed if any of the model assumptions appear to be violated. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Not applicable.

## 2.2. Study Objective(s) and Endpoint(s)

| Ob | jectives | En | dpoints |
|---|---|---|---|
| | Part 1 | | |
| Pri | mary Objectives | Pri | imary Endpoints |
| • | To investigate the safety and tolerability of GSK3342830 after administration of single IV doses in healthy adult subjects | • | Clinical safety data from AEs, clinical laboratory tests, vital signs (blood pressure, heart rate, temperature, and respiration rate), and 12-lead ECG readings |
| Se | condary Objectives | Pri | imary Objectives |
| • | To determine the pharmacokinetics of GSK3342830 after administration of single IV doses in healthy adult subjects | • | Plasma and urine concentrations PK endpoints include AUC(0-t), AUC(0-∞), Cmax, Tmax, CL, Vss, t1/2, Feu(t1-t2), Ae, and CLr of GSK3342830, as data permit |
| • | To assess dose proportionality of GSK3342830 after administration of single IV doses in healthy adult subjects | • | Pharmacokinetic endpoints include AUC(0-t), AUC(0-∞), and Cmax of GSK3342830 after administration of single IV doses for the assessment of dose proportionality, as data permit |
| Ex | ploratory Objectives | Ex | ploratory Endpoints |
| • | To correlate PK parameters (AUC[0-t], AUC[0-∞], and Cmax) of GSK3342830 with safety findings after administration of single IV doses in healthy adult subjects | • | Exposure-response analyses, as data permit |
| • | To evaluate the production of any GSK3342830 metabolites in plasma and urine and determine the need to perform a more detailed analysis of any metabolites | • | Metabolite characterization in plasma and urine and estimation of observed drug-related material in plasma to determine the presence of any metabolite >10%, and estimate the percentage dose eliminated via urine |
| | Par | | = |
| Pri | mary Objectives | Pri | imary Endpoints |
| • | To investigate the safety and tolerability of GSK3342830 after administration of repeat IV doses in healthy adult subjects | • | Clinical safety data from AEs, clinical laboratory tests, vital signs (blood pressure, heart rate, temperature, and respiration rate), and 12-lead ECG readings |
| Secondary Objectives | | Se | condary Endpoints |
| • | To determine the pharmacokinetics of GSK3342830 after administration of repeat IV doses in healthy adult subjects | • | Plasma and urine concentrations and PK endpoints include AUC(0-t) and AUC(0- $\infty$ ) on Day 1 only, AUC(0- $\tau$ ), Cmax, Tmax, CL, Vss, t1/2, C $\tau$ , Feu(t1- t2), Ae, and CLr of GSK3342830, as data permit |
| • | To assess dose proportionality of GSK3342830 after administration of repeat IV doses in healthy adult subjects | • | Pharmacokinetic endpoints include AUC(0- $\tau$ ) and Cmax of GSK3342830 after administration of repeat IV doses for the assessment of dose proportionality, as data permit |

| Oh | jectives | En | dpoints |
|---|---|---|---|
| • | To examine the extent of accumulation, time invariance, and achievement of steady-state of GSK3342830 after administration of repeat IV doses in healthy adult subjects | • | Observed accumulation ratio (Ro) based on AUC and Cmax of GSK3342830 after administration of repeat IV doses, as data permit Steady-state ratio (Rss) of GSK3342830 to assess time invariance, as data permit Trough plasma concentrations at the end of the dosing interval ( $C\tau$ ) to assess the achievement of steady-state of GSK3342830 after administration of repeat IV doses, as data permit |
| Ex | ploratory Objectives | Ex | ploratory Endpoints |
| • | To correlate PK parameters (AUC[0-t], AUC[0-∞], AUC[0-τ], and Cmax) of GSK3342830 with safety findings in healthy adult subjects after administration of repeat IV doses | • | Exposure-response analyses, as data permit |
| • | To evaluate the production of any GSK3342830 metabolites in plasma and urine and determine the need to perform a more detailed analysis of any metabolites | • | Metabolite characterization in plasma and urine and estimation of observed drug-related material in plasma to determine the presence of any metabolite >10%, and estimate the percentage dose eliminated via urine |
| | Par | | |
| Pri | mary Objectives | Pri | mary Endpoints |
| • | To investigate the safety and tolerability of GSK3342830 after administration of a single IV dose in healthy adult Japanese subjects | • | Clinical safety data from AEs, clinical laboratory tests, vital signs (blood pressure, heart rate, temperature, and respiration rate), and 12-lead ECG readings |
| Se | condary Objectives | Se | condary Endpoints |
| • | To determine the pharmacokinetics of GSK3342830 after administration of a single IV dose in healthy adult Japanese subjects | • | Plasma and urine concentrations PK endpoints include AUC(0-t), AUC(0-∞), Cmax, Tmax, CL, Vss, t1/2, Feu(t1-t2), Ae, and CLr of GSK3342830, as data permit |
| Ex | ploratory Objectives | Ex | ploratory Endpoints |
| • | To correlate PK parameters (AUC[0-t], AUC[0-∞], and Cmax) of GSK3342830 with safety findings in healthy adult Japanese subjects after administration of repeat IV doses | • | Exposure-response analyses, as data permit |
| • | To evaluate the production of any GSK3342830 metabolites in plasma and urine and determine the need to perform a more detailed analysis of any metabolites | • | Metabolite characterization in plasma and urine and estimation of observed drug-related material in plasma to determine the presence of any metabolite >10%, and estimate the percentage dose eliminated via urine |

## 2.3. Study Design



Note: Figure shows illustration of the planned doses, which may be switched, changed, or cancelled based on preliminary safety, tolerability, and pharmacokinetic data from preceding cohorts.

Part 2 Repeat Dose Escalation Study Design Schematic



Note: Figure shows illustration of the planned doses, which may be switched, changed, or cancelled based on preliminary safety, tolerability, and pharmacokinetic data from preceding cohorts.

#### Design Features

- Part 1 is planned to include 6 dose level cohorts. Up to 2 additional doses (1 per cohort) may be evaluated to further understand the study drug. The planned starting GSK3342830 dose in Part 1 is 250 mg administered as a single IV infusion. The dose is planned to increase in subsequent cohorts to 500, 1000, 2000, 4000, and ≤6000 mg IV.
  - In Part 1, subjects will remain confined to the clinical unit from admission on Day –1 until all scheduled safety and PK assessments have been completed on Day 3. The duration of study (from Screening to the Follow-up visit) for each subject will be up to approximately 43 days.
- Part 2 is planned to include a sequential panel of up to 3 dose level cohorts.
   Additional repeat dose cohorts may be evaluated to further assess the safety, tolerability, and pharmacokinetics of GSK3342830. The planned starting GSK3342830 dose in Part 2 is 1000 mg administered as a single IV infusion on Day 1, TID IV infusions on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14, and a single IV infusion on Day 15. The dose is planned to increase in subsequent cohorts to 2000 and 4000 mg TID.
  - In Part 2, subjects will remain confined to the clinical unit from admission on Day –1 until after all scheduled safety assessments have been completed on Day 16. The duration of study (from Screening to the Follow-up visit) for each subject will be up to approximately 56 days.
- Part 3 is planned to include 1 cohort (Cohort J). The planned GSK3342830 dose in Part 3 will be either 250, 500, 1000, 2000, 4000, or \$6000 mg based on preliminary safety and tolerability results of doses determined to be safe and well tolerated in subjects of non-Japanese heritage after completion of the single escalation dose cohorts (Part 1). The dose in Part 3 will be

| Overview of S | tudy Design and Key Features |
|---|---|
| | administered as a single IV infusion on Day 1. |
| | In Part 3, subjects will remain confined to the clinical unit from admission on |
| | Day –1 until all scheduled safety and PK assessments have been completed on Day 3. The duration of study (from Screening to the Follow-up visit) for |
| | each subject will be up to approximately 43 days. |
| Dosing | <ul> <li>For Part 1, doses are planned to escalate in a sequential fashion contingent<br/>on the safety, tolerability, and PK profile of approximately 4 subjects who<br/>received active treatment in the previous cohort. The evaluated subjects<br/>should be followed for a minimum of 48 hours after dosing. Dose escalations</li> </ul> |
| | or reductions will progress with modifications based on the preliminary safety, tolerability, and PK data from the preceding cohorts. |
| | <ul> <li>For Part 2, doses are planned to escalate in a sequential fashion based on the preliminary safety, tolerability, and PK data from Part 1 and at least 14 days of repeat dosing in approximately 5 subjects who received active treatment in the previous cohort in Part 2. The evaluated subjects should be followed for a minimum of 24 hours after dosing on Day 15. The dosing frequency, duration</li> </ul> |
| | of dosing, and decision to dose in the next dose level may be changed based on the safety, tolerability, or PK findings in Part 1 or earlier doses in Part 2. |
| | The dose in Part 3 will be administered as a single IV infusion on Day 1. |
| Treatment Assignment | <ul> <li>For Part 1 on Day 1, before study drug administration, subjects will be<br/>randomized to treatment with either GSK3342830 or placebo in a 3:1 ratio. As</li> </ul> |
| Assignment | a safety precaution, all Part 1 cohorts will be split into 2 sub-cohorts for |
| | sentinel dosing. In each cohort, the first 2 subjects will receive either |
| | GSK3342830 or placebo (1 active/1 placebo). Dosing in the remaining 6 |
| | subjects (5 active/1 placebo) in that cohort will occur at least 24 hours later |
| | <ul> <li>based on the safety results from the first sub-cohort.</li> <li>For Part 2 on Day 1, before study drug administration, subjects will be</li> </ul> |
| | randomized to treatment with either GSK3342830 or placebo in a 4:1 ratio. |
| | <ul> <li>For Part 3 on Day 1, before study drug administration, subjects will be</li> </ul> |
| Into vivo | randomized to treatment with either GSK3342830 or placebo in a 4:1 ratio. |
| Interim<br>Analysis | <ul> <li>No formal interim analysis. However, during dose escalation, Bayesian<br/>analysis is performed to produce inferences about model parameters and the</li> </ul> |
| Allalysis | predictive probability that an individual will have certain PK parameters larger |
| | than prespecified thresholds at for each dose level to aid the next dose |
| | selection. |

## 2.4. Statistical Hypotheses

No inferential hypothesis testing will be performed.

#### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No formal interim analysis is planned for this study. However, one may be conducted in the event of clinically significant safety or PK findings. All preliminary safety, tolerability, and available PK data will be reviewed internally at GSK and with the clinical study site before each dose escalation in Part 1, before initiation of Part 2, and before each dose escalation in Part 2.

The relationship between dose and plasma GSK3342830 exposure, and associated variability will be characterized by a power model once data are available from 3 dose levels. Prior to that, prediction of the human exposure at the next dose will be based on population PK modeling (if feasible) or on the assumption of dose–exposure proportionality (i.e., doubling the dose gives an approximate doubling of exposure). If prior PK results show less than proportional increase in exposure with increasing dose, the prediction will be based on the assumption that the fold exposure increase to fold dose increase ratio will be the same with the current dose escalation as it was with the previous one. If prior PK results show more than proportional increase in exposure with dose, subsequent dose escalations will not be higher than 3-fold. The power model will be updated as data become available throughout the study. During dose escalation, Bayesian inferential probability that a group mean will have AUCs (AUC[0-t] for single dose and AUC[0-8]x3 as AUC[0-24] for repeat dose) and Cmax values greater than 2875 h•μg/mL and 2270 μg/mL (mean exposures at the NOAEL dose in the rat and monkey), respectively, and Bayesian predictive probability that an individual will have AUC(0-24) and Cmax values greater than 3460 houg/mL and 2590 ug/mL (maximum exposures at the NOAEL dose in the rat for AUC and the monkey for Cmax), respectively, may be calculated for the next dose level and used together with safety and tolerability data to aid the next dose selection.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to PPD procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Safety | Defined as all subjects who receive at least 1 dose of study drug and have at least 1 post-dose safety assessment. | <ul><li>Study Population</li><li>Safety</li></ul> |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | This population will be based on the treatment<br>the subject was randomized to receive. | |
| Pharmacokinetic | Defined as all subjects who receive at least 1 dose of GSK3342830 and have evaluable PK data for GSK3342830. | • PK |
| Pharmacokinetic<br>Parameter | Defined as all subjects in the PK population for<br>whom valid and evaluable PK parameters<br>were derived | PK Parameter |

#### NOTES:

• Please refer to Appendix 11: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Time & Events |
| 10.2 | Appendix 2: Treatment States and Phases |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| 10.6 | Appendix 6: Values of Potential Clinical Importance |
| 10.6 | Appendix 7: DMID Adult Toxicity Tables for Adverse Event Assessment |
| 10.8 | Appendix 8: Multiple Comparisons & Multiplicity |
| 10.9 | Appendix 9: Model Checking and Diagnostics for Statistical Analyses. |
| 10.10 | Appendix 10: Abbreviations & Trade Marks. |
| 10.11 | Appendix 11: List of Data Displays. |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data | Displays Gene | rated |
|---|---|---|---|
| | Table | Figure | Listing |
| Randomisation | | | |
| Randomisation | | | Υ |
| Subject Disposition | | | |
| Subject Disposition | Υ | | Υ |
| Reason for Screening Failures | Υ | | Υ |
| Reason for Withdrawals | Υ | | Υ |
| Inclusion and Exclusion Criteria Deviations | | | Υ |
| Demography | | | |
| Demographic Characteristics | Υ | | Υ |
| Medical Conditions and Concomitant Medications | | | |
| Concomitant Medication | Y | | Υ |
| Medical Conditions (Current/Past) | Y | | Y |

NOTES:

Y = Yes display generated.

## 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Safety Analyses

## 7.1.1. Overview of Planned Safety Analyses

The safety analyses will be based on the Safety population, unless otherwise specified.

Table 3 provides an overview of the planned Safety analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 3 Overview of Planned Safety Analyses

| Display Type | | Abs | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sun | nmary | Indiv | ridual | Sum | mary | Individual | |
| | Т | F | F | L | T | F | F | L |
| Exposure | | | | | | | | |
| Extent of Exposure | Υ | | | Υ | | | | 1 |
| Adverse Events | | | | | | | | |
| All AEs | Y | | | Υ | | | | 1 |
| All Drug-Related AEs | Y | | | Υ | | | | · |
| Serious AEs | | | | Υ | | | | |
| Withdrawal AEs | | | | Υ | | | | |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry | Υ | | | Υ | Υ | | | |
| Hematology | Υ | | | Υ | Υ | | | |
| Urinalysis (Dipstick) | Υ | | | Υ | | | | |
| ECGs | | | | | | | | |
| ECG Findings | Υ | | | Υ | | | | |
| ECG Values | Υ | | | Υ | Υ | | | |
| Vital Signs | | | | | | | | |
| Vital Signs | Y | | | Υ | Υ | | | · |
| Cardiac Telemetry | | | | | | | | |
| Cardiac Telemetry | | | | Υ | | | | · |
| Liver | | | | | | | | |
| Liver Events [1] | | | | Υ | | | | |
| Cardiovascular | | | | | | | | |
| Cardiovascular Events | | | | Υ | | | | i |
| [1] | | | | | | | | |
| Injection Site Reactions | 6 | | | | | | | |
| Injection Site Reaction | | | | Υ | | | | · |
| Events [1] | | | | | | | | |
| Rash | | | | | | | | |
| Rash Events [1] | | | | Υ | | | | 1 |
| Biomarker | | | | | | | | |
| Cytokines | | | Υ | Υ | | | | <u> </u> |

#### CONFIDENTIAL

204847

#### NOTES:

- 1. Conditional displays, they will only be produced when an event has occurred.
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents TFL related to any displays of individual subject observed raw data.

#### 8. SECONDARY STATISTICAL ANALYSES

## 8.1. Pharmacokinetic Analyses

## 8.1.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the PK population, unless otherwise specified.

Table 4 provides an overview of the planned PK analyses, with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 4 Overview of Planned Pharmacokinetic Analyses

| Endpoint / | | | Un | transf | ormed | | | Log-Transformed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stat | s Analy | ysis | Sun | nmary | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Indiv | idual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| PK Plasma | | | | V | <b>Y</b> [1] [2] | <b>Y</b> [1] | V | | | | | | | |
| Concentrations | | | | ī | 11.11. | 11.1 | I | | | | | | | |
| PK Urine | | | | | | | V | | | | | | | |
| Concentrations | | | | | | | ľ | | | | | | | |
| PK Plasma | V | | | V | | V | V | V | | | V | | | |
| Parameters | ı | | | ī | | ī | I | I | | | ī | | | |
| PK Urine | | | | V | | V | V | | | | | | | |
| Parameters | | | | ĭ | | T | ľ | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Linear and Semi-Log plots will be created on the same display.
- [2] Separate mean, median, and median trough (Part 2 only) concentration plots will be generated.

## 8.1.2. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).

#### 8.1.3. Pharmacokinetic Parameters

#### 8.1.3.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher.

- All calculations of non-compartmental parameters will be based on actual sampling times.
- Pharmacokinetic parameters described in Table 5 will be determined from the plasma GSK3342830 concentration-time data, as data permits.
- Pharmacokinetic parameters described in Table 6 will be determined from the urinary GSK3342830 concentration data, as data permits.

Table 5 Derived Plasma Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| Cmax | Maximum plasma concentration |
| Tmax | Time to Cmax |
| AUC(0-t) | AUC from time zero to the last quantifiable concentration after dosing |
| AUC(0-∞) | AUC extrapolated from time 0 to infinity (estimated for single dose in Part 1 and Part 3 and on Day 1 for repeat dose in Part 2) |
| AUC(0-τ) | AUC over the dosing interval $\tau$ |
| t1/2 | Terminal elimination half-life |
| CL | Total systemic clearance |
| Vss | Steady-state volume of distribution |
| Сτ | Trough concentration |
| Ratio of invariance | Time invariance ratio, calculated by (AUC(0- $\tau$ ) on Day 15)/(AUC(0- $\infty$ ) on Day 1) |
| Ratio of accumulation | Accumulation ratio, calculated by $(AUC(0-\tau) \text{ on Day } 15)/(AUC(0-\tau) \text{ on Day } 1)$ |

#### NOTES:

Additional parameters may be included as required.

Table 6 Derived Urinary Pharmacokinetic Parameters

| Parameter | Parameter Description |
|------------|------------------------------------------|
| Feu(t1-t2) | Urinary excretion ratio relative to dose |
| CLr | Renal clearance |
| Ae | Amount excreted in urine |

#### 8.1.3.2. Statistical Analysis of Pharmacokinetic Parameters

The following pharmacokinetic statistical analyses will only be performed, if sufficient data is available (i.e. if subjects have well defined plasma profiles).

| Pharmacokinetic Statistical Analyses |
|--------------------------------------|
| Assessment |
| Dose proportionality of GSK3342830. |

#### **Pharmacokinetic Statistical Analyses**

#### Endpoint(s)

• An estimate of slope (with corresponding 90% CI).

#### **Model Specification**

 Dose proportionality of AUC(0-∞) and Cmax on Day 1 after single dose (Part 1) and for repeat dose groups (Day 15 in Part 2), AUC(0-τ) and Cmax of GSK3342830 on Day 15 will be assessed separately by day using the following power model:

$$y = \alpha * dose^{\beta}$$
.

where y denotes the PK parameter being analyzed and  $\alpha$  depends on the random error in the repeat dose phase where subjects take the study drug in a parallel-group fashion. Dose proportionality implies that  $\beta$ =1 and will be assessed by estimating  $\beta$  along with its 90% CI. The exponent,  $\beta$ , in the power model will be estimated by regressing the loge-transformed PK parameter on loge-transformed dose.

$$log(y) = log(\alpha) + \beta * log(dose)$$

The power model will be fitted by restricted maximum likelihood (REML) using Statistical Analysis Software (SAS) Proc Mixed, with a fixed effect term for dose. The PK parameter endpoint and the factor dose will be loge-transformed prior to the analysis.

• In the case where dose proportionality is not established over the entire dosing range, secondary analysis of dose proportionality will be assessed for select doses over the higher dosing range with the power model or by pair-wise analysis of variance (ANOVA) using the SAS mixed models procedure. If the secondary analysis using the pair-wise ANOVA approach is performed, a reference dose would be chosen based on the lowest clinically relevant dose over which the pharmacokinetics can be adequately described and the other doses would be treated as test doses.

## **Model Checking & Diagnostics**

Refer to Appendix 9: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

 An estimate of slope (with corresponding 90% CI) will be provided as a measure of potential dose proportionality (i.e. a slope of approximately 1 implies dose proportionality) will be produced in tabular format.

#### **Assessment**

• Time invariance of GSK3342830.

#### Endpoint(s)

• An estimate of time invariance ratio (with corresponding 90% CI).

#### **Model Specification**

For the repeat dose cohorts (Part 2), the time invariance ratio will be assessed by fitting a mixed effect model for  $AUC(0-\infty)$  on Day 1 and  $AUC(0-\tau)$  on Day 15 data with subject as a random effect and group (group=1 for  $AUC(0-\infty)$  on Day 1, and group=2 for  $AUC(0-\tau)$  on Day 15) as a fixed effect for each cohort.

### **Model Checking & Diagnostics**

Refer to Appendix 9: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

• The time invariance ratio of GSK3342830 will be estimated by calculating the ratio of the geometric least squares means of group 1 (AUC(0- $\tau$ ) on Day 15) to group 2 (AUC(0- $\infty$ ) on Day 1) and the corresponding 90% CI for each cohort.

#### Assessment

#### **Pharmacokinetic Statistical Analyses**

Accumulation ratio of GSK3342830.

#### Endpoint(s)

• An estimate of accumulation ratio (with corresponding 90% CI).

#### **Model Specification**

• For the repeat dose cohorts (Part 2), the accumulation ratio (Ro) will be calculated as the ratio of AUC(0-τ) on Day 15 to AUC(0-τ) on Day 1 for each subject. The dosing interval (τ) will be equal to 8 hours. Following log-transformation, AUC(0-τ) of GSK3342830 on Days 1 and 15 will be analyzed by a mixed effect model, fitting dose, day, and dose-by-day interaction as fixed effects and subject as a random effect. For each dose, point estimate and 90% CI for the difference "AUC(0-τ) on Day 15 - AUC(0-τ) on Day 1" will be constructed using the appropriate error term. The point estimate and associated 90% CI will then be exponentially backtransformed to provide point and 90% CI estimates for the ratios "AUC(0-τ) on Day 1." If dose-by-day interaction is not significant, then a single point estimate and 90% CI pooled across all doses for the ratio AUC(0-τ) on Day 15: AUC(0-τ) on Day 1 may be constructed with all estimates for each dose.

### **Model Checking & Diagnostics**

Refer to Appendix 9: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

• The point estimate and 90% CI for the accumulation ratios of AUC(0- $\tau$ ) on Day 15 to AUC(0- $\tau$ ) on Day 1 will be calculated.

#### Assessment

Steady state assessment of GSK3342830.

#### Endpoint(s)

• An estimate of the slope (with corresponding 90% CI).

#### **Model Specification**

• To evaluate whether steady state was achieved, statistical analysis of steady-state  $C_{\tau}$  will be performed after log-transformation of  $C_{\tau}$  on Days 3, 6, 9, 12, 13, and 15. A mixed effect model will be fitted by dose and day (as a continuous covariate) as a fixed effect term and subject as a random effect term. Distributional assumptions underlying the statistical analyses will be assessed by visual inspection of residual plots. Normality will be examined by normal probability plots, while homogeneity of variance will be assessed by plotting the residuals against the predicted values for the model. Alternative analyses of the data will be performed if any of the model assumptions appear to be violated.

#### **Model Checking & Diagnostics**

• Refer to Appendix 9: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

 The coefficients for the slope of the day effect on the log-scale will be used to evaluate steadystate for each dose group. Using the pooled estimate of variance, the 90% CIs for the slope will be calculated.

#### **Model Results Presentation**

 The least squares geometric mean ratio and 90% CI for the comparison of AUC(0-t), AUC(0-∞) and Cmax from Japanese subjects (Part 3) to subjects of non-Japanese heritage of the same dose level (Part 1) will be calculated.

#### **Assessment**

Assessment of GSK3342830 PK in healthy adult Japanese subjects vs the same dose level of

## Pharmacokinetic Statistical Analyses

healthy adult subjects in Part 1.

### Endpoint(s)

• The geometric mean ratio and associated 90% CI for Part 3 vs Part 1.

## Model Specification

• To evaluate whether there is a difference in the PK parameters in healthy adult Japanese subjects, a fixed effect model will be fitted with Study Part as fixed effect.

## **Model Checking & Diagnostics**

• Refer to Appendix 9: Model Checking and Diagnostics for Statistical Analyses.

## **Model Results Presentation**

• The geometric mean ratio and associated 90% CI will be presented in a table.

### 8.2. Bayesian Dose Escalation Analyses

#### 8.2.1. Overview of Planned Bayesian Dose Escalation Analyses

The Bayesian Dose Escalation analyses will be based on the PK population, unless otherwise specified.

Table 7 provides an overview of the planned Bayesian analyses, with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 7 Overview of Planned Bayesian Analyses

| Endpoint / | | Untransformed | | | | | Log-Transformed | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stat | s Anal | ysis | Sun | nmary | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Indiv | idual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| AUC[0-t],<br>AUC[0-24],<br>AUC[0-8]x3,<br>Cmax | | | | Y | Y | | Y | Y | Υ | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data, posterior distribution data and predictive data about future hypothetical subjects.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 8.2.2. Planned Bayesian Statistical Analyses

#### Table 8 Bayesian Statistical Analyses

#### **Bayesian Statistical Analyses**

#### Endpoint(s)

- AUC[0-t] where t varies depending dose and Cmax for Part 1 single dose phase
- AUC[0-24] which is calculated as AUC[0-8]x3, Cmax for Part 2 repeat dose phase

#### **Model Specification**

To guide dose selection, Bayesian posterior inferences about population probability distributions of model parameters of PK parameters will be assessed by using the following power model:

$$y = \exp(\theta_1 + \varepsilon) \cdot dose^{\theta_2}$$

where y denotes the PK parameter being analyzed. The  $\theta_s$ , s=1,2, in the power model will be estimated by linear regression of the loge-transformed PK parameters on loge dose levels.

$$\log(y_{ij}) = \theta_1 + \theta_2 \cdot \log(d_{ij}) + \varepsilon_{ij} \tag{1}$$

where

- y<sub>tf</sub> is the observed or predicted log-PK variable of the j-th dose d<sub>ij</sub> administered to the i-th subject. In particular, it is an AUC (AUC[0-t] for single dose, and AUC[0-24] for repeat dose) or a Cmax, as applicable.
- \$\mathcal{G}\_{\mathcal

#### **Bayesian Statistical Analyses**

•  $\epsilon_{ij}$  is a random error term, with mean zero and variance  $\sigma^2$ .

In general, Bayesian inference seeks to quantify the probability distributions of model parameters such as the  $(\theta_1, \theta_2, \sigma)$  defined in Equation (1). The present inference will incorporate a normal-Half-Normal prior distribution, to express the prior information about the parameters  $(\theta_1, \theta_2, \sigma)$ . Due to limited information available about the GSK3342830 compound, an informative prior with large variance will be used. For ease of parameterization for the normal distribution in computer programming, use  $v = \sigma^{-2}$  as the precision. Model parameters are assumed a priori to be independent.

Table 9 Prior Distributions

| Model Parameter | Prior |
|---|---|
| <b>0</b> ₁ (intercept) | ~ Normal(-1, precision=10-6)* |
| $\theta_{_{Z}}$ (slope of log-dose) | ~ Half-Normal(0, precision=10 <sup>-5</sup> , lower=0)* |
| ₩ (precision) | ~ Gamma(1, iscale=5)* |

All model parameters are a prioiri independent.

\*SAS Version 9.4 will be used for the Bayesian analysis, specifying the normal distribution using mean and precision. Because of the assumption that population mean PK parameter values increase as a higher dose is administered, let  $\theta_2$  have a Half Normal prior distribution truncated at 0 to guarantee the positivity of  $\theta_2$ . Simple linear regression, with maximum likelihood estimation, on available data at dose escalation will be used to estimate the model parameters ( $\theta_1, \theta_2, \nu$ ), thus providing the initial values for model parameter estimation by Bayesian approach; however, if insufficient data are available for estimation, (1, -1, 0.2) will be used as the initial values for  $(\theta_1, \theta_2, \nu)$ . Furthermore, the scale and shape parameters of the precision prior Gamma function are chosen to attain  $E(\nu)=0.2$  and  $Var(\nu)=0.04$ . Two chains will be run for the estimation of each parameter.

## **Model Checking & Diagnostics**

The Gibbs sampling chains will be run using the following conventions:

- 1. The burn-in period, the number of iterations judged necessary for the Markov Chain Monte Carlo (MCMC) algorithm to achieve convergence, will be assessed after each 5,000 iteration increment until convergence is achieved. Convergence of the chains to the posterior distribution will be assessed using:
- Gelman-Rubin statistic
- MCMC error of the chains
- Autocorrelation plot to assess autocorrelation within each chain
- Visual inspection of the chain trace plots for proper chain mixing after the application of thinning
- 2. The burn-in samples must meet all the following convergence criteria, before we accept

#### **Bayesian Statistical Analyses**

the MCMC output as a sample from the posterior distribution:

- 1) The Gelman-Rubin statistic will indicate convergence provided the Brooks-Gelman Ratio (Brooks and Gelman 1998) for all parameters is within the interval (0.8, 1.2). The SAS procedure diagnostic tool will generate the necessary output.
- 2) All MCMC chains will be run until each parameter has estimated MCMC error of less than 5% of its associated standard deviation. This calculation will be performed as the ratio of the MCMC error divided by the parameter's estimated posterior standard deviation.
- 3) Autocorrelation plots will be generated for all chains and accepted provided the estimated autocorrelation for each chain is within  $\pm 0.10$  by lag 10. In the event that any chain's autocorrelations for any one parameter are outside that range after 10 iterations, the number of iterations will be increased by 5000.
- 4) All chains' trace plots will be inspected visually, to assess the mixing of each chain. Convergence is indicated when all chains appear to be mixing well (to be clear: No chain's convergence is indicated until the chains of all model parameters appear well-mixed). Mixing is defined as "each chain is sampling independently values similar to those the other chains have sampled." This will appear in the trace plots as all chains overlapping each other randomly.

The burn-in period will end at the iteration which convergence is reached as determined using the above criteria. Upon convergence a sample size of 10,000 will be obtained from the posterior from each chain. Estimated density plots will be created and inspected for smoothness. If the estimated density plots are not smooth, then an additional sample size of 10,000 iterations, 10,000 from each chain, will be gathered until the estimated density plots are smooth. Estimates for each parameter will include mean, standard deviation, MCMC error, median, and the centred 90% credible sets (the 5th and 95th percentiles) along with the estimated MCMC error for the chain. We will also obtain the Deviance Information Criteria for the model and display this with the associated output.

Poor fit for the model will be indicated by the following, possibly among other findings:

- 1) Patterns in the residuals.
- 2) The model requires more than 10,000 iterations for the burn-in period, after thinning, and an acceptable reparameterisation of the model is not found or it is determined that the chains will not reach convergence.

#### **Model Results Presentation**

Once the posterior distributions have been estimated using SAS, the following key interim analysis inferences and predictions will be estimated using the associated posteriors:

Univariate features of the posterior probability distribution (mean, StdDev, MCMC error, ratio of MCMC error/StdDev, median, and 5<sup>th</sup> and 95<sup>th</sup> percentiles used for 90% equaltailed credible intervals (CrI)) will be calculated for each model parameter. The estimated dose response curve with a 90% CrI will be graphically displayed, and overlaid on the

#### **Bayesian Statistical Analyses**

observed data.

- The range of possible doses: 250, 500, 1000, 2000, 4000 and 6000 mg for Part 1 and 1000, 2000, 4000 mg for Part 2.
- At each chain of the MCMC algorithm in the SAS program (as described above), we will obtain an estimate for the mean AUC[0-t] or Cmax at each dosing level (as in the previous bullet for Part 1) with a 90% CrI using the 5<sup>th</sup> and 95<sup>th</sup> percentiles. This will be calculated as found in the model formulation (1) using the sampled parameter values.
- These point estimates will be displayed on a figure with the dots connected. If the associated posterior distributions for the predicted responses at the dose levels are skewed then the point estimates used to generate the dose response curve plot will be generated using the median as a measure of central tendency. The 5<sup>th</sup> and 95<sup>th</sup> percentiles will still be used for the 90% CrI about the parameter.
- The observed data will be overlaid on this curve at the doses which were explored.
- The Bayesian inferential probability that mean AUC[0-t] and Cmax values will be greater than 2875 h.μg/mL and 2270 μg/mL (maximum exposures at the NOAEL dose in the rat for AUC and the monkey for Cmax), respectively, will be calculated for each dose level in Part 1.
- The Bayesian predictive probability that an individual subject will have AUC[0-t] and Cmax values greater than 3460 h.μg/mL and 2590 μg/mL (maximum exposures at the NOAEL dose in the rat for AUC and the monkey for Cmax), respectively, will be calculated for each dose level in Part 1.

All the outputs discussed above and listed below are used together with safety and tolerability data to aid the next dose selection.

The mean, median, and 5<sup>th</sup> and 95<sup>th</sup> percentiles (90% CrI) for each model parameter and prediction will be tabulated.

Figures will be produced for posterior dose-response model for AUC[0-t], and Cmax (with 90% Crl), respectively as discussed above in inference bullet.

A Listing for PK parameters AUC[0-t] and Cmax in Part I single dose phase will be provided.

In addition, the above listed inferences and predictions will be performed for PK parameters AUC[0-24] and Cmax in Part 2 repeat dose phase. The corresponding tables, figure and listing listed above will also be produced.

#### Sensitivity and Supportive Statistical Analyses

Not applicable.

## 8.2.3. Deviations from RAP Planned Analysis

To ensure transparency, any deviations from the above analyses will be documented in a log appended to the CSR. These deviations may include (although are not limited to) algebraically different model parameterizations or changes in the prior structure to support convergence of the parameter estimations in SAS. These possible issues and solutions for them are discussed above in the appropriate sections.

## 9. REFERENCES

GlaxoSmithKline Document Number 2015N257523\_01 (Amendment 1 – 01-NOV-2016): A Phase I, Randomized, Double-Blind (Sponsor Unblinded), Single-Center, Placebo-Controlled, Three-Part Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Ascending Single and Repeat Intravenous Doses of GSK3342830 in Healthy Adult Subjects.

## 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.1 | Appendix 1: Time and Events |
| Section 10.2 | Appendix 2: Treatment States & Phases |
| Section 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.4 | Appendix 4: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| | Pharmacokinetic |
| | Pharmacodynamic and or Biomarkers |
| Section 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.6 | Appendix 6: Values of Potential Clinical Importance |
| Section 10.8 | Appendix 7: DMID Adult Toxicity Tables for Adverse Event Assessment |
| Section 10.8 | Appendix 8: Multiple Comparisons and Multiplicity |
| Section 10.9 | Appendix 9: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 10.10 | Appendix 10: Abbreviations & Trade Marks |
| Section 10.11 | Appendix 11: List of Data Displays |

## 10.1. Appendix 1: Time & Events

## 10.1.1. Protocol Defined Time & Events

## Time and Events Table: Screening and Day –1; Single and Repeat Dose Escalation (Part 1 and Part 2) and Single Dose (Part 3)

| Procedure | Screening (up to 30 days before Day 1) | Day -1 | Notes |
|---|---|---|---|
| Informed consent | Χ | | |
| Inclusion and exclusion criteria | X | Χ | |
| Demography | X | | |
| Medical history (includes substance usage and family history of premature cardiovascular disease) | Х | Х | Substances: drugs, alcohol, tobacco and caffeine. |
| Past and current medical conditions including cardiovascular medical history | X | Х | |
| Safety and Laboratory Assessments | | | |
| SAE review | Х | Х | Serious AEs will be collected from the signing of informed consent. |
| Concomitant medication review | Х | Х | |
| Full physical examination including height and weight | X | | |
| Brief physical examination | | Χ | |
| Vital signs (BP, HR, oral temperature, respiration rate) | Χ | Х | |
| 12-lead electrocardiogram | X | Х | |
| Continuous cardiac monitoring | | Х | Continuous dual-lead telemetry will be initiated on Day –1 at least 8 hours before study drug administration on Day 1. |
| Urine cotinine and drug and breath alcohol screens | Χ | Χ | |
| β-hCG pregnancy test/estradiol/FSH | Х | Х | Pregnancy test (if female of child-bearing age; serum at screening and urine at Day –1); estradiol and FSH at screening as appropriate. Only women of non-child-bearing potential may participate. |
| Human immunodeficiency virus antibody, hepatitis B surface antigen, and hepatitis C antibody screen | X | | |
| Table is continued on the next page. | | | |

| Procedure | Screening (up to 30 days before Day 1) | Day -1 | Notes |
|---|---|---|---|
| Clinical chemistry (including liver chemistries), hematology, and urinalysis | X | х | The albumin to creatinine ratio will be determined at Screening using the first morning void urine as described in protocol Section 7.3.7. An aliquot of the urine sample will be collected for NGAL and KIM-1 at Day –1. These samples may be analyzed after the end of the study if a clinical signal is detected. Instructions for collection and storage of these urine samples are included in the Study Reference Manual. Hematology assessments on Day –1 will also include total iron, total binding iron capacity, ferritin, and reticulocytes. |
| Genetic sample | | Х | Collect a pharmacogenomics sample only if the subject has a signed consent specific for this purpose. The pharmacogenomics sample can be collected anytime, but Day –1 is recommended. Informed consent for optional sub-studies (e.g., genetics research) must be obtained before collecting a sample. |
| Admission to clinical unit | | Х | |

β-hCG = beta human chorionic gonadotropin, BP = blood pressure, FSH = follicle-stimulating hormone, HR = heart rate, KIM-1 = kidney injury molecule 1, NGAL = neutrophil gelatinase-associated lipocalin, SAE = serious adverse event.

#### Time and Events Table: Part 1 - Single Dose Escalation and Part 3 - Single Dose

| | Day 1 | | | | | | | | | | | | | Da | ıy 2 | Day 3 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Hours relative to treatment administration | | | | | | | | | | | | | | | | | | | |
| | Pre-dose | 0 | 0.5 | 1 | 1.25 | 1.5 | 2 | 3 | 3.5 | 4 | 4.5 | 5 | 6 | 8 | 10 | 12 | 16 | 24 | 36 | 48 |
| Randomization | Χ | | | | | | | | | | | | | | | | | | | |
| 12-lead ECG <sup>1</sup> | Χ | | Χ | Χ | | Χ | Χ | Χ | | Χ | | | Χ | | | Χ | | Χ | | Х |
| Vital signs (BP, HR, oral temperature, respiration rate) | Χ | | Х | Χ | | Х | Χ | Х | | Х | | | Х | | | Х | | Χ | | Х |
| Fasting clinical chemistry,<br>hematology, and urinalysis <sup>2</sup> | | | | | | | | | | | | | | | | | | Χ | | |
| Treatment administration <sup>3</sup> | | Χ | | | | | | | | | | | | | | | | | | i |
| Blood collection for pharmacokinetics <sup>4</sup> | Χ | | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Χ | Χ | Χ | Х |
| Urine collection for pharmacokinetics5 | X | X | | | | | | | | X | | | | X | | X | | X- | | X |
| Continuous cardiac monitoring <sup>6</sup> | Χ← | | | | | | Co | ntinuo | ıs revie | :W | | | | | | | | | | <del></del> |
| AE review | XContinuous review | | | | | | | <del>→</del> | | | | | | | | | | | | |
| SAE review | X← | | | | | | | | | | | | | | | | | | | |
| Concomitant medication review | X | X← | | | | | | | <del>→</del> | | | | | | | | | | | |
| Discharge from inpatient unit <sup>7</sup> | | | | | | | | | | | | | | | | | | | | Х |

AE = adverse event, BP = blood pressure, ECG = electrocardiogram, HR = heart rate, SAE = serious adverse event. NOTES:

- 1. Triplicate 12-lead ECGs to be obtained at least 5 minutes apart within 1 hour before dosing. Single ECGs will be obtained at all other time points.
- 2. An aliquot of the urine sample will be collected for neutrophil gelatinase-associated lipocalin (NGAL) and kidney injury molecule 1 (KIM-1). These samples may be analyzed after the end of the study if a clinical signal is detected. Instructions for collection and storage of these urine samples are included in the Study Reference Manual. The albumin to creatinine ratio will be determined using the first morning void urine on Day 2.
- 3. GSK3342830 or placebo will be administered as a single IV infusion in the morning on Day 1. The planned infusion duration time is 1 hour.
- 4. Pharmacokinetic blood samples will be collected for GSK3342830 and potential metabolites. At the end of the study the saved blood samples from a predicted therapeutically-relevant dose level and higher dose level for plasma PK analysis of parent and the highest dose level completed for metabolite profile, will be transferred to a GSK specified laboratory. Details of PK sample collection and storage will be provided in the Study Reference Manual.
- 5. Pooled urine samples will be collected over the following time intervals: pre-dose (within a 24-hour period before dosing, may begin on Day –1) and 0 to 4, 4 to 8, 8 to 12, 12 to 24, and 24 to 48 hours post-dose. Two aliquots of urine samples for baseline analysis may be collected from any time after admission to just before dosing on Day 1. At the end of the study, the saved urine samples from a predicted therapeutically-relevant dose level and higher dose level for urinary PK analysis of parent and the highest dose level completed for potential metabolite profile, will be transferred to a GSK specified laboratory. Urine will be collected in opaque bottles to maintain blind of blinded study site personnel. Details of urine sample collection and storage will be provided in the Study Reference Manual.
- 6. Continuous dual-lead telemetry will be initiated on Day –1 at least 8 hours before treatment administration on Day 1 and will continue until 48 hours post dose.
- 7. Subjects will be discharged from the clinical unit after the 48-hour post-dose assessments are complete.

#### Time and Events Table: Part 2 - Repeat Dose Escalation

| Dropoduro | | Study Day | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| Randomization | Х | | | | | | | | | | | | | | | |
| 12-lead ECG <sup>1</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Vital signs (BP, HR, oral temperature, respiration rate) <sup>2</sup> | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Fasting clinical chemistry, hematology, and urinalysis tests <sup>3</sup> | | Х | | | Х | | | | | Х | | | | | Х | |
| Treatment administration <sup>4</sup> | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Χ | Х | Χ | Х | |
| Blood collection for pharmacokinetics <sup>5</sup> | Х | | Х | | | Х | | | Х | | | Χ | Х | | Х | |
| Urine collection for pharmacokinetics <sup>6</sup> | Χ | Χ | | | | | | | | | | | | | Χ | Χ |
| Continuous cardiac monitoring <sup>7</sup> | X←Cor | ntinuous r | eview→ | | | | | | | | | | | | | |
| AE review | X <del>←</del> | | | | | | -Continu | ous revie | W | | | | | | | · |
| SAE review | XContinuous review | | | | | | <del></del> | | | | | | | | | |
| Concomitant medication review X | | | | | | | Continu | ous revie | W | | | | | | | <del>-</del> |
| Discharge from inpatient unit <sup>8</sup> | | | | | | | | | | | | | | | | Х |

AE = adverse event, BP = blood pressure, ECG = electrocardiogram, HR = heart rate, SAE = serious adverse event. NOTES:

- 1. Triplicate 12-lead ECGs will be obtained at least 5 minutes apart within 1 hour before the start of infusion (pre-dose) on Day 1. Single ECGs will be obtained at 0.5, 1, 1.5, 2, 3, 4, 6, and 12 hours after the start of infusion on Day 1 and Day 15, within 1 hour before the start of the morning infusion on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14, and in the morning on Day 16.
- 2. Vital signs will be measured within 1 hour before the start of infusion (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, and 12 hours after the start of infusion on Days 1 and 15, within 1 hour before the start of the morning infusion and on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14, and in the morning on Day 16.
- 3. An aliquot of the urine sample will be collected for neutrophil gelatinase-associated lipocalin (NGAL) and kidney injury molecule 1 (KIM-1). These samples may be analyzed after the end of the study if a clinical signal is detected. Instructions for collection and storage of these urine samples are included in the Study Reference Manual. Hematology assessments on Days 5 and 15 will also include total iron, total iron binding capacity, ferritin, and reticulocytes. The albumin to creatinine ratio will be determined using the first morning void urine on Days 5 and 15.
- 4. GSK3342830 or placebo will be administered as a single IV infusion in the morning on Day 1, TID IV infusions (approximately every 8 hours) on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14, and as a single IV infusion in the morning on Day 15. The planned infusion duration time is 1 hour.

Footnotes are continued on the next page.

#### CONFIDENTIAL

#### 204847

- 5. Pharmacokinetic samples for GSK3342830 and potential metabolites will be collected on Day 1 at the following time points: pre-dose (within 15 minutes before dosing) and 0.5, 1 (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hours after the start of infusion. Single pre-dose trough samples will be taken on the mornings of Days 3, 6, 9, 12, and 13. Serial samples will be collected on Day 15 at the following time points: pre-dose (within 15 minutes before dosing) and 0.5, 1 (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after the start of infusion. At the end of the study, the saved blood samples from a predicted therapeutically-relevant dose level and higher dose level for plasma PK analysis of parent and from the highest dose level completed for potential metabolite profile will be transferred to a GSK specified laboratory. Details of PK sample collection and storage will be provided in the Study Reference Manual.
- 6. Pooled urine samples will be collected on Day 1 and Day 15 over the following time intervals: pre-dose (within a 24-hour period before dosing, may begin on Day –1) and 0 to 8 and 8 to 24 hours post-dose. Two aliquots of urine samples for baseline analysis may be collected from any time after admission to just before dosing on Day 1. At the end of the study, the saved urine samples from a predicted therapeutically-relevant dose level and higher dose level for urinary PK analysis of parent and from the highest dose-level completed for potential metabolite profile, will be transferred to a GSK specified laboratory. Urine will be collected in opaque bottles to maintain blind of blinded study site personnel. Details of urine sample collection and storage will be provided in the Study Reference Manual.
- 7. Continuous dual-lead telemetry will be initiated on Day –1 at least 8 hours before treatment administration on Day 1 and will continue until 48 hours post dose.
- 8. Subjects will be discharged from the clinical unit after the Day 16 assessments are complete.

#### Time and Events Table: Follow-up Visit; Single and Repeat Dose Escalation (Part 1 and Part 2) and Single Dose (Part 3)

| Procedure | Follow-up Visit (7 to 10 days post last dose or early termination) |
|---|---|
| Adverse event/serious adverse event review | X |
| Concomitant medication review | X |
| Brief physical examination | X |
| 12-lead electrocardiogram | Х |
| Vital signs | Х |
| Urine β-human chorionic gonadotropin pregnancy test (women of child-bearing age) | X |
| Clinical chemistry, hematology, and urinalysis tests <sup>1</sup> | X |

#### NOTE:

<sup>1.</sup> An aliquot of the urine sample will be collected for neutrophil gelatinase-associated lipocalin (NGAL) and kidney injury molecule 1 (KIM-1). These samples may be analyzed after the end of the study if a clinical signal is detected. Instructions for collection and storage of these urine samples are included in the Study Reference Manual. Hematology assessments will also include total iron, total iron binding capacity, ferritin, and reticulocytes. The albumin to creatinine ratio will be determined using the first morning void urine as described in protocol Section 7.3.7.

## 10.2. Appendix 2: Treatment States and Phases

#### 10.2.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to dosing.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date |
| Post-Treatment | Date > Study Treatment Stop Date |

#### 10.2.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

## 10.2.2.1. Treatment States for Safety Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date/time < Study Treatment Start Date/time |
| On-Treatment | Study Treatment Start Date/time ≤ Date/time ≤ Study Treatment Stop Date/time + 2 days |
| Post-Treatment | Date/time > Study Treatment Stop Date/time + 2 days |

#### NOTES:

• If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

#### 10.2.2.2. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date/time < Study Treatment Start Date/time |
| On-Treatment | If AE onset date/time is on or after treatment start date & on or before treatment stop date/time. |
| | Study Treatment Start Date/time ≤ AE Start Date/time ≤ Study Treatment Stop Date/time + 2 days |
| Post-Treatment | If AE onset date/time is after the treatment stop date/time. |
| | AE Start Date/time > Study Treatment Stop Date/time + 2 days |
| Onset Time<br>Since 1st Dose | If Treatment Start Date/time > AE Onset Date/time, = AE Onset Date - Treatment Start Date |
| (Days) | If Treatment Start Date/time ≤ AE Onset Date/time, = AE Onset Date - Treatment Start Date +1 |
| | Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on CRF OR value is missing. |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

### 10.3.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | | |
|---|---|---|---|---|
| | Ran | domization Schedule | Data Displays for Repor | ting |
| Part | Code | Description | Description | Order [1] |
| 1 | A1 | Cohort A GSK3342830 | GSK3342830 250 mg | 1 |
| 1 | A2 | Cohort B GSK3342830 | GSK3342830 500 mg | 2 |
| 1 | A3 | Cohort C GSK3342830 | GSK3342830 1000 mg | 3 |
| 1 | A4 | Cohort D GSK3342830 | GSK3342830 2000 mg | 4 |
| 1 | A5 | Cohort E GSK3342830 | GSK3342830 4000 mg | 5 |
| 1 | A6 | Cohort F GSK3342830 | GSK3342830 6000 mg | 6 |
| 1 | A7 | Cohort X1 GSK3342830 | GSK3342830 XXXX <sup>[3]</sup> mg | 7 |
| 1 | A8 | Cohort X2 GSK3342830 | GSK3342830 XXXX <sup>[3]</sup> mg | 8 |
| 1 | Р | Placebo | Placebo | 9 |
| 2 | A9 | Cohort G GSK3342830 | GSK3342830 1000 mg TID | 10 |
| 2 | A10 | Cohort H GSK3342830 | GSK3342830 2000 mg TID | 11 |
| 2 | A11 | Cohort I GSK3342830 | GSK3342830 4000 mg TID | 12 |
| 2 | A12 | Cohort Y1 GSK3342830 | GSK3342830 XXXX <sup>[3]</sup> mg TID | 13 |
| 2 | A13 | Cohort Y2 GSK3342830 | GSK3342830 XXXX <sup>[3]</sup> mg TID | 14 |
| 2 | Р | Placebo | Placebo | 15 |
| 3 | AJ1 | Cohort J GSK3342830 | GSK3342830 XXXX <sup>[4]</sup> mg | 16 |
| 3 | PJ | Placebo | Placebo | 17 |
| 3 | AJ2 | Cohort Z1 GSK3342830 | GSK3342830 XXXX <sup>[4]</sup> mg | 18 |
| 3 | PJ | Placebo | Placebo | 19 |

#### NOTES:

- 1. Order represents treatments being presented in TFL, as appropriate.
- 2. Cohort X1, X2, Y1, and Y2 are created per protocol to allow 2 additional doses which may be evaluated to further understand the study drug. The Randomization Schedule does not contain the actual dose levels but instead refers to the Cohort dose level. Dose levels may change from the protocol defined levels. The TLFs will display the actual dose levels used in the study.
- 3. The dose for Cohort X1, X2, Y1, and Y2 will be determined once the decision is made to enroll those optional cohorts.
- 4. The dose for Cohort J will either 250, 500, 1000, 2000, 4000 or ≤6000 mg based on preliminary safety and tolerability results of doses determined to be safe and well tolerated in subjects of non-Japanese heritage after completion of the single escalation dose cohorts (Part 1).
#### 10.3.2. Baseline Definition & Derivations

#### 10.3.2.1. Baseline Definitions

For all endpoints (expect as noted in baseline definitions) the baseline value will be the latest pre-dose assessment.

| Parameter | Study Assess | Baseline Used in | | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety | Safety | | | |
| Hematology | Х | Χ | | Day -1 |
| Clinical Chemistry | Х | Χ | | Day -1 |
| 12 Lead ECG | Х | Χ | X | Day 1 (Pre-dose) |
| Vital Signs | Х | Χ | Х | Day 1 (Pre-dose) |

#### NOTES:

 Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

# 10.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.3.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

## 10.3.3. Reporting Process & Standards

# Reporting Process

#### Software

 The currently supported versions of SAS software [Insert Other Software as Required] will be used.

#### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.1.3 & AdaM IG Version 1.0.
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

# **Generation of RTF Files**

RTF files will be generated for all reporting efforts described in the RAP.

# Reporting Standards

#### General

## **Reporting Standards**

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - o 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| 7 ill disolicatica visits will be included in listings. | |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharm | acokinetic Concentration Data |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharmacokinetic Parameters | |
| Descriptive<br>Summary Statistics<br>(Log Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CVb- (%)) will be reported. |
| (Log Transionnieu) | CV <sub>b</sub> (%) = $\sqrt{(\exp(SD^2) - 1) * 100}$<br>(SD = SD of log transformed data) |

# **CONFIDENTIAL**

| Reporting Standards | |
|---|---|
| Parameters Not<br>Being Log<br>Transformed | Tmax, %AUCex, tlast, lambda_z, lambda_z_lower, lambda_z_upper, lambda_z_no. of points, Ratio of time invariance, Ratio of accumulation, Feu(t1-t2), CLr, Ae |
| Listings | Include all following PK parameters: Cmax, AUC0- $\infty$ , AUC0-t, AUC(0- $\tau$ ), t1/2, CL, Vss, C $\tau$ , Ratio of time invariance, Ratio of accumulation, Tmax, %AUCex, tlast, lambda_z, lambda_z_lower, lambda_z_upper, lambda_z_no. of points, Feu(t1-t2), CLr, Ae. |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# **Reporting Standards**

# 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. General

# **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

# **Study Day**

- Calculated as the number of days from treatment date :
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < Treatment Date → Study Day = Ref Date Treatment Date</li>
- Ref Data ≥ Treatment Date → Study Day = Ref Date (Treatment Date) + 1

# 10.4.2. Study Population

## **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>

# 10.4.3. Safety

#### **ECG Parameters**

#### **RR** Interval

- IF ECG values are machine read and RR interval (msec) is not provided directly, then RR interval can be derived as:
  - [1] If QTcB is machine read & RR is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and RR is not provided, then:

# **ECG Parameters**

$$RR = \left[ \left( \frac{QT}{QT cF} \right)^2 \right] * 1000$$

- If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.
- Important Note: Machine read values of RR should not be replaced with re-derived values.

# **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

 Important Note: Machine read values of QTcB and QTcF should not be replaced with re-derived values. If neither machine read QTcB or QTcF are available but QT and RR are collected, then a QTcB and QTcF can be derived however this should be discussed and agreed with the study team and the TLFs must have an appropriate footnote denoting those parameters are derived.

#### **Adverse Events**

# **AE'S OF Special Interest**

- Liver events
- CV events
- Infusion site reactions
- Potential systemic allergic reactions
- Hematologic events
- Rash Events

# 10.5. Appendix 5: Premature Withdrawals and Handling of Missing Data

# 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as one who has completed all phases of the study including the follow-up visit.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.5.2.1. Handling of Missing Dates

| Reporting Detail |
|---|
| Partial dates will be displayed as captured in subject listing displays. |
| <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 2: Treatment States and Phases.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be</li> </ul> |
| F |

| Element | Reporting Detail |
|---|---|
| | Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied. |

# 10.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

| Advorce | Any model dates for advance counts will be united to date group against If the |
|---|---|
| Adverse | Any partial dates for adverse events will be raised to data management. If the |
| Events | full date cannot be ascertained, the following assumptions will be made: |
| | o If the partial date is a start date, a '01' will be used for the day and 'Jan' will |
| | be used for the month. |
| | <ul> <li>However, if these results in a date prior to Week 1 Day 1 and the event</li> </ul> |
| | could possibly have occurred during treatment from the partial information, |
| | then the Week 1 Day 1 date will be assumed to be the start date. |
| | <ul> <li>The AE will then be considered to start on-treatment (worst case).</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day</li> </ul> |
| | (dependent on the month and year) and 'Dec' will be used for the month. |
| | The recorded partial date will be displayed in listings. |

# 10.6. Appendix 6: Values of Potential Clinical Importance

# 10.6.1. ECG

| ECG Parameter | Units | Potential Clinical Importance Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| | | > 450 [1] | |
| Abasista OTs Interval | msec | > 450 [2] | ≤ 479 <sup>[2]</sup> |
| Absolute QTc Interval | | ≥ 480[2] | ≤ 499 <sup>[2]</sup> |
| | | ≥ 500 <sup>[2]</sup> | |
| Absolute PR Interval | msec | < 110 <sup>[1]</sup> | > 220 [1] |
| Absolute QRS Interval | msec | < 75 [1] | > 110 [1] |
| Change from Baseline | | | |
| | msec | <b>≤30</b> [2] | |
| Increase from Baseline QTc | msec | > 30[2] | ≤ 59 <sup>[2]</sup> |
| | msec | ≥ 60 <sup>[1]</sup> | |

# NOTES:

- 1. Represent standard ECG values of PCI for HV studies.
- 2. Represent further subdivisions of ECG values for analysis.

# 10.6.2. Vital Signs

| Vital Sign Parameter | Units | Potential Clinical Importance Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 10.7. Appendix 7: DMID Adult Toxicity Tables for Adverse Event Assessment

# 10.7.1. Laboratory Values

Parameter values are converted to use SI units.

# HEMATOLOGY

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hemoglobin | 95 to 105 G/L | 80 to 94 G/L | 65 to 79 G/L | <65 G/L |
| Absolute neutrophil count | 1.0 to 1.5 10^9/L | 0.75 to 0.999 10^9/L | 0.5 to 0.749 10^9/L | <0.5 10^9/L |
| Platelets | 75 to 99.999 10^9/L | 50 to 74.999 10^9/L | 20 to 49.999 10^9/L | <20 10^9/L |
| White Blood Cells | 11 to 13 10^9/L | 13 to 15 10^9/L | 15 to 30 10^9/L | >30 or <1 10^9/L |
| % Polymorphonuclear leukocytes + band cells | >80% | 90 to 95% | >95% | N/A |
| Abnormal Fibrinogen | Low: 1 to 2 G/L<br>High: 4 to 6 G/L | Low: <1 G/L<br>High: >6 G/L | Low: <0.5 G/L<br>High: N/A | Fibrinogen associated with gross bleeding or with disseminated coagulation |
| Fibrin Split Product | 0.020 to 0.040 G/L | 0.041 to 0.050 G/L | 0.051 to 0.060 G/L | >0.060 G/L |
| Prothrombin Time | 1.01 to 1.25 × ULN | 1.26 to 1.5 × ULN | 1.51 to 3.0 × ULN | >3 × ULN |
| Activated Partial Thromboplastin | 1.01 to 1.66 × ULN | 1.67 to 2.33 × ULN | 2.34 to 3 × ULN | >3 × ULN |
| Methemoglobin | 5.0 to 9.9% | 10.0 to 14.9% | 15.0 to 19.9% | >20% |

N/A = not applicable; ULN = upper limit of normal.

#### CHEMISTRIES

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hyponatremia | 130 to 135 MMOL/L | 123 to 129 MMOL/L | 116 to 122 MMOL/L | <116 MMOL/L or abnormal sodium with mental status changes or seizures |
| Hypernatremia | 146 to 150 MMOL/L | 151 to 157 MMOL/L | 158 to 165 MMOL/L | >165 MMOL/L or abnormal sodium with mental status changes or seizures |
| Hypokalemia | 3.0 to 3.4 MMOL/L | 2.5 to 2.9 MMOL/L | 2.0 to 2.4 MMOL/L or intensive replacement therapy of hospitalization required | <2.0 MMOL/L or abnormal potassium with paresis, ileus, or life-threatening arrhythmia |
| Hyperkalemia | 5.6 to 6.0 MMOL/L | 6.1 to 6.5 MMOL/L | 6.6 to 7.0 MMOL/L | >7.0 MMOL/L or abnormal potassium with |

| | | | | life threatening arrhythmia |
|---|---|---|---|---|
| | | | | life-threatening arrhythmia <1.67 MMOL/L or abnormal glucose with |
| Hypoglycemia | 3.0 to 3.55 MMOL/L | 2.22 to 2.99 MMOL/L | 1.67 to 2.21 MMOL/L | mental status changes or coma |
| Hyperglycemia<br>(nonfasting and no prior<br>diabetes) | 6.44 to 8.88 MMOL/L | 8.89 to 13.88 MMOL/L | 13.89 to 27.75 MMOL/L | >27.76 MMOL/L or abnormal glucose with ketoacidosis or seizures |
| Hypocalcemia (corrected for albumin) | 2.10 to 1.95 MMOL/L | 1.94 to 1.75 MMOL/L | 1.74 to 1.52 MMOL/L | <1.52 MMOL/L or abnormal calcium with life-threatening arrhythmia or tetany |
| Hypercalcemia (corrected for albumin) | 2.64 to 2.87 MMOL/L | 2.88 to 3.12 | 3.13 to 3.37 MMOL/L | >3.37 MMOL/L or abnormal calcium with life-threatening arrhythmia |
| Hypomagnesemia | 0.7 to 0.6 MMOL/L | 0.59 to 0.45 MMOL/L | 0.44 to 0.3 MMOL/L | <0.3 MMOL/L or abnormal magnesium with life-threatening arrhythmia |
| Hypophosphatemia | 0.7 to 0.8 MMOL/L | 0.5 to 0.6 MMOL/L or replacement Rx required | 0.3 to 0.4 MMOL/L intensive therapy or hospitalization required | <0.3 MMOL/L or abnormal phosphate with life-threatening arrhythmia |
| Hyperbilirubinemia (when accompanied by any increase in other liver function test) | 1.1 to <1.25 × ULN | 1.25 to <1.5 × ULN | 1.5 to 1.75 × ULN | >1.75 × ULN |
| Hyperbilirubinemia (when other liver function tests are in the normal range) | 1.1 to <1.5 × ULN | 1.5 to <2.0 × ULN | 2.0 to 3.0 × ULN | >3.0 × ULN |
| Blood urea nitrogen | 1.25 to 2.5 × ULN | 2.6 to 5 × ULN | 5.1 to 10 × ULN | >10 × ULN |
| Hyperuricemia (uric acid) | 446 to 595 UMOL/L | 596 to 714 UMOL/L | 715 to 892 UMOL/L | >892 UMOL/L |
| Creatinine | 1.1 to 1.5 × ULN | 1.6 to 3.0 × ULN | 3.1 to 6.0 × ULN | >6 × ULN or dialysis required |

Rx = therapy; ULN = upper limit of normal.

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Aspartate aminotransferase | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Alanine aminotransferase | $1.1 \text{ to } < 2.0 \times \text{ ULN}$ | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Gamma to glutamyl transferase | $1.1 \text{ to } < 2.0 \times \text{ ULN}$ | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Alkaline Phosphatase | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Amylase | 1.1 to 1.5 × ULN | 1.6 to 2.0 × ULN | 2.1 to 5.0 × ULN | >5.1 × ULN |
| Lipase | 1.1 to 1.5 × ULN | 1.6 to 2.0 × ULN | 2.1 to 5.0 × ULN | >5.1 × ULN |

ULN = upper limit of normal.

| URINALYSIS | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Drotoinurio | 1+ or | 2 to 3+ or | 4+ or | Nephrotic syndrome or |
| Proteinuria | 200 MG to 1 GM loss/day | 1 to 2 GM loss/day | 2 to 3.5 GM loss/day | >3.5 GM loss/day |
| Homoturio | Microscopic only | Gross, no clots | Gross, with or without clots, | Obstructive or |
| Hematuria | <10 RBC/HPF | >10 RBC/HPF | or red blood cells casts | required transfusion |

HPF = high-powered field; RBC = red blood cells.

# 10.8. Appendix 8: Multiple Comparisons & Multiplicity

# 10.8.1. Handling of Multiple Comparisons & Multiplicity

No adjustments for multiplicity will be made.

# 10.9. Appendix 9: Model Checking and Diagnostics for Statistical Analyses

# 10.9.1. Statistical Analysis Assumptions

| Endpoint(s) | • | PK endpoints AUC and Cmax |
|-------------|---|---------------------------|
| Analysis | • | Mixed Effects |

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- Distributional assumptions underlying the statistical analyses will be assessed by visual inspection of residual plots. Normality will be examined by normal probability plots, while homogeneity of variance will be assessed by plotting the residuals against the predicted values for the model.

# 10.10. Appendix 10 – Abbreviations & Trade Marks

# 10.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| Ae | Amount excreted in urine |
| AUC | Area under the curve |
| AUC(0-t) | AUC from time zero to the time of last quantifiable concentration |
| $AUC(0-\infty)$ | AUC from time zero to infinity |
| AUC(0-τ) | AUC over the dosing interval τ |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CL | Total systemic clearance |
| CLr | Renal clearance |
| Cmax | Concentration at maximum |
| Сτ | Trough concentration |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CrI | Credible interval |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> /CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| Feu(t1-t2) | Urinary excretion ratio relative to dose |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| GUI | Guidance |
| MCMC | Markov Chain Monte Carlo |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |

| Abbreviation | Description |
|---|---|
| Ratio of | Accumulation ratio, calculated by AUC(0- $\tau$ ) on day 15/ AUC(0- $\tau$ ) on |
| accumulation | day 1 |
| Ratio of time | Time invariance ratio, calculated by AUC(0- $\tau$ ) on day 15/ AUC(0- $\infty$ ) on |
| invariance | day 1 |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| t1/2 | Terminal elimination half-life |
| Tmax | Time of maximum concentration |
| Vss | Steady-state volume of distribution |
| GSK | GlaxoSmithKline |

# 10.10.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| WinNonlin |
| SAS |

# 10.11. Appendix 11: List of Data Displays

# 10.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables Figures | |
|------------------|------------------------|-----|
| Study Population | 1.1 to 1.9 | |
| Safety | 2.1 to 2.17 | 2.1 |
| Pharmacokinetic | 3.1 to 3.22 3.1 to 3.2 | |
| Section | Listings | |
| ICH Listings | 1 to 47 | |

# 10.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in the TLF Specification documents.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 10.11.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| DE [X] | Dose Escalation |
| SAC [X] | Final Statistical Analysis Complete |

# NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 10.11.4. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition a | nd Analysis Sets | | | |
| 1.1 | Safety | NS | Summary of Number of Subjects Enrolled by Country and Site ID | | SAC [1] |
| 1.2 | Safety | ES1 | Summary of Subject Disposition | | SAC [1] |
| 1.3 | Screened | ES6 | Summary of Reasons for Screening Failures | | SAC [1] |
| 1.4 | Screened | DV1 | Summary of Important Protocol Deviations | | SAC [1] |
| Demog | raphics and Ba | seline Characteri | stics | | · |
| 1.5 | Safety | DM1 | Summary of Demographic Characteristics | | SAC [1] |
| 1.6 | Safety | DM11 | Summary of Age Ranges | | SAC [1] |
| 1.7 | Safety | DM5 | Summary of Race and Racial Combinations | | SAC [1] |
| 1.8 | Safety | DM6 | Summary of Race and Racial Combinations Details | | SAC [1] |
| Medica | I Conditions | | | · | <u> </u> |
| 1.9 | Safety | MH1 | Summary of Cardiovascular Related Medical Conditions | | SAC [1] |

# 10.11.5. Safety Tables

| Safet | y : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Adve | rse Events | | | | • |
| 2.1 | Safety | AE2 | Relationship of Adverse Event System Organ Classes, Preferred Terms and Verbatim Text | | SAC [1] |
| 2.2 | Safety | AE1 | Summary of All Adverse Events | | SAC [1] |
| 2.3 | Safety | AE1 | Summary of Drug-Related Adverse Events | | SAC [1] |
| 2.4 | Safety | A15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC [1] |
| 2.5 | Safety | A16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC [1] |
| Labo | ratory Measur | ements | | • | • |
| 2.6 | Safety | LB1 | Summary of Clinical Chemistry Values | | SAC [1] |
| 2.7 | Safety | LB1 | Summary of Clinical Chemistry Change from Baseline | | SAC [1] |
| 2.8 | Safety | LB1 | Summary of Haematology Values | | SAC [1] |
| 2.9 | Safety | LB1 | Summary of Haematology Change from Baseline | | SAC [1] |
| 2.10 | Safety | UR3b | Summary of Urinalysis Dipstick Results | | SAC [1] |
| Elect | rocardiogram | S | | | |
| 2.11 | Safety | EG1 | Summary of ECG Findings | | SAC [1] |
| 2.12 | Safety | EG2 | Summary of ECG Values | | SAC [1] |
| 2.13 | Safety | EG2 | Summary of Change from Baseline in ECG Values | | SAC [1] |
| 2.14 | Safety | SAFE_T1 | Summary of Frequency of Maximum Post-Dose ECG Parameter Corrected QTc Interval | | SAC [1] |

| Safet | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.15 | Safety | SAFE_T2 | Summary of Frequency of Maximum Change from Baseline for ECG Parameter Corrected QTc Interval | | SAC [1] |
| Vital | Vital Signs | | | | |
| 2.16 | Safety | VS1 | Summary of Vital Signs | | SAC [1] |
| 2.17 | Safety | VS1 | Summary of Vital Signs Change from Baseline | | SAC [1] |

# 10.11.6. Safety Figures

| Safety : Fig | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Cytokine Pl | ots | | | | |
| 2.1 | Safety | SAFE_F1 | Boxplot of Cytokine Data | | SAC [1] |
| 2.2 | Safety | SAFE_F2 | Individual Cytokine Plot | | SAC [1] |

# 10.11.7. Pharmacokinetic Tables

| Pharmacol | kinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Concer | ntration Data | | | | |
| 3.01 | PK | PK01 | Summary of GSK3342830 Single Dose Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment in Part 1 and Part 3 | | SAC [1] |
| 3.02 | PK | PK01 | Summary of GSK3342830 Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment in Part 2 | | SAC [1] |
| PK Parame | eters | | | | |
| 3.03 | PK Parameter | PKPT1 | Summary of Untransformed GSK3342830 Single Dose Plasma Pharmacokinetic Parameters in Part 1 and Part 3 | Tmax, %AUCex, tlast, lambda_z, lambda_z_lower, lambda_z_upper, lambda_z_no. of points | SAC [1] |
| 3.04 | PK Parameter | PKPT3 | Summary of Log-transformed GSK3342830 Single Dose Plasma Pharmacokinetic Parameters in Part 1 and Part 3 | Cmax, AUC(0-t), AUC(0-∞), t1/2, CL, Vss | SAC [1] |
| 3.05 | PK Parameter | PKPT1 | Summary of Untransformed GSK3342830 Single Dose Urine Pharmacokinetic Parameters in Part 1 and Part 3 | Feu(t1-t2), CLr, Ae | SAC [1] |
| 3.06 | PK Parameter | PKPT1 | Summary of Untransformed GSK3342830 Plasma<br>Pharmacokinetic Parameters in Part 2 | Cmax, AUC(0-t), AUC(0-∞), AUC(0-τ), t1/2, CL, Vss, Cτ, Ratio of time invariance, Ratio of accumulation, Tmax, %AUCex, tlast, lambda_z, lambda_z_lower, lambda_z_upper, lambda_z_no. of points | SAC [1] |
| 3.07 | PK Parameter | PKPT3 | Summary of Log-transformed GSK3342830 Plasma Pharmacokinetic Parameters in Part 2 | Cmax, AUC(0-t), AUC(0-∞), AUC(0-τ), t1/2, CL, Vss, Cτ | SAC [1] |

| Pharmaco | kinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.08 | PK Parameter | PKPT1 | Summary of Untransformed GSK3342830 Urine Pharmacokinetic Parameters in Part 2 | Feu(t1-t2), CLr, Ae | SAC [1] |
| PK Analys | is Tables | • | | | |
| 3.09 | PK Parameter | PK_T1 | Summary of Statistical Analysis of GSK3342830 Plasma Dose Proportionality in Part 1 | Cmax, AUC(0-∞) | SAC [1] |
| 3.10 | PK Parameter | PK_T1 | Summary of Statistical Analysis of GSK3342830 Plasma Dose Proportionality in Part 2 | Cmax, AUC(0-τ) | SAC [1] |
| 3.11 | PK Parameter | PK_T1 | Summary of Statistical Analysis of GSK3342830 Plasma Time Invariance in Part 2 | AUC(0-∞) on Day 1 and AUC(0-τ) on Day 15 | SAC [1] |
| 3.12 | PK Parameter | PK_T1 | Summary of Statistical Analysis of GSK3342830 Plasma<br>Accumulation Ratio in Part 2 | AUC(0-τ) | SAC [1] |
| 3.13 | PK Parameter | PK_T1 | Summary of Statistical Analysis of GSK3342830 Plasma Steady State Assessment in Part 2 | Cτ | SAC [1] |
| Bayesian I | Dose Escalation | • | | | |
| 3.14 | PK Parameter | PK_T2 | Summary of Model Parameters for Part 1 - Posterior Distributions | | DE [1] |
| 3.15 | PK Parameter | PK_T2 | Summary of Model Parameters for Part 2 - Posterior Distributions | | DE [1] |
| 3.16 | PK Parameter | PK_T3 | Summary of PK Parameters for Part 1 - Bayesian Prediction of Individual Subjects | | DE [1] |
| 3.17 | PK Parameter | PK_T3 | Summary of PK Parameters for Part 2 - Bayesian Prediction of Individual Subjects | | DE [1] |
| 3.18 | PK Parameter | PK_T4 | Summary of PK Parameters for Part 1 - Bayesian Predictive Probability | | DE [1] |

| Pharmacol | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.19 | PK Parameter | PK_T4 | Summary of PK Parameters for Part 2 - Bayesian Predictive Probability | | DE [1] |
| 3.20 | PK Parameter | PK_T4 | Summary of PK Parameters for Part 1 - Bayesian Inferential Probability | | DE [1] |
| 3.21 | PK Parameter | PK_T4 | Summary of PK Parameters for Part 2 - Bayesian Inferential Probability | | DE [1] |
| 3.22 | PK Parameter | PK_T1 | Summary of Statistical Analysis of GSK3342830 Single Dose Plasma Pharmacokinetic Parameters in Part 1 and Part 3 Subjects | | SAC [1] |

# 10.11.8. Pharmacokinetic Figures

| harmacok | inetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Concentrat | ion Plots | | | | 1 |
| 3.01 | PK | PKCF4 | Mean (SD) GSK3342830 Single Dose Plasma Concentration-<br>Planned Time Plots for Part 1 and Part 3 (Linear and Semi-<br>Log) | | SAC [1] |
| 3.02 | PK | PKCF5 | Median (range) GSK3342830 Single Dose Plasma<br>Concentration-Planned Time Plots for Part 1 and Part 3 (Linear<br>and Semi-Log) | | SAC [1] |
| 3.03 | PK | PKCF4 | Mean (SD) GSK3342830 Plasma Concentration-Planned Time Plots for Part 2 (Linear and Semi-Log) | | SAC [1] |
| 3.04 | PK | PKCF5 | Median (range) GSK3342830 Plasma Concentration-Planned Time Plots for Part 2 (Linear and Semi-Log) | | SAC [1] |
| 3.05 | PK | PKCF5 | Median (range) GSK3342830 Plasma Pre-dose Concentration versus Day for Part 2 (Linear and Semi-Log) | | SAC [1] |
| 3.06 | PK | PKCF1P | Individual GSK3342830 Single Dose Plasma Concentration-<br>Planned Time Plots for Part 1 and Part 3 (Linear and Semi-Log) | | SAC [1] |
| 3.07 | PK | PKCF1P | Individual GSK3342830 Plasma Concentration-Planned Time Plots for Part 2 (Linear and Semi-Log) | | SAC [1] |
| PK Parame | ters | | | | |
| 3.08 | PK Parameter | PKPF3 | Comparative Plot of Individual GSK3342830 Plasma AUC(0-t) Versus Dose for Part 1 | | SAC [1] |
| 3.09 | PK Parameter | PKPF3 | Comparative Plot of Individual GSK3342830 Plasma AUCinf Versus Dose for Part 1 | | SAC [1] |

| Pharmacol | kinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10 | PK Parameter | PKPF3 | Comparative Plot of Individual GSK3342830 Plasma Cmax Versus Dose for Part 1 | | SAC [1] |
| 3.11 | PK Parameter | PKPF3 | Comparative Plot of Individual GSK3342830 Plasma Ae Versus Dose for Part 1 | | SAC [1] |
| 3.12 | PK Parameter | PKPF3 | Comparative Plot of Individual GSK3342830 Plasma AUC(0-t) Versus Dose on Day 1 for Part 2 | | SAC [1] |
| 3.13 | PK Parameter | PKPF3 | Comparative Plot of Individual GSK3342830 Plasma AUC(0-∞) Versus Dose on Day 1 for Part 2 | | SAC [1] |
| 3.14 | PK Parameter | PKPF3 | Comparative Plot of Individual GSK3342830 Plasma Cmax Versus Dose on Day 1 for Part 2 | | SAC [1] |
| 3.15 | PK Parameter | PKPF3 | Comparative Plot of Individual GSK3342830 Plasma Ae Versus Dose on Day 1 for Part 2 | | SAC [1] |
| 3.16 | PK Parameter | PKPF3 | Comparative Plot of Individual GSK3342830 Plasma AUCtau Versus Dose on Day 15 for Part 2 | | SAC [1] |
| 3.17 | PK Parameter | PKPF3 | Comparative Plot of Individual GSK3342830 Plasma Cmax<br>Versus Dose on Day 15 for Part 2 | | SAC [1] |
| 3.18 | PK Parameter | PKPF3 | Comparative Plot of Individual GSK3342830 Plasma Ae Versus Dose on Day 15 for Part 2 | | SAC [1] |
| Bayesian [ | Dose Escalation | | | <u> </u> | |
| 3.19 | PK Parameter | PK_F1 | AUC[0-t] (µg.h/mL) in Part 1 - Dose Response Curve | | DE [1] |
| 3.20 | PK Parameter | PK_F1 | Cmax (µg/mL) in Part 1 - Dose Response Curve | | DE [1] |
| 3.21 | PK Parameter | PK_F1 | AUC[0-24] (µg.h/mL) in Part 2 - Dose Response Curve | | DE [1] |
| 3.22 | PK Parameter | PK_F1 | Cmax (µg/mL) in Part 2 - Dose Response Curve | | DE [1] |

# **10.11.9. ICH Listings**

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Rando | misation | , | | | |
| 1 | Safety | TA1 | Listing of Randomized and Actual Treatments | | SAC [1] |
| Subjec | ct Disposition | | | | |
| 2 | Safety | ES2 | Listing of Reasons for Study Withdrawal | | SAC [1] |
| 3 | Screened | ES7 | Listing of Reasons for Screening Failure | | SAC [1] |
| 4 | Screened | DV2 | Listing of Important Protocol Deviations | | SAC [1] |
| 5 | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC [1] |
| Demo | graphics | | | | |
| 6 | Safety | DM2 | Listing of Demographic Characteristics | Include height, weight,<br>BMI, Smoking History,<br>Alcohol History,<br>Caffeine History, and<br>Drug Use History | SAC [1] |
| 7 | Safety | DM9 | Listing of Race | | SAC [1] |
| Medic | al Conditions and | Concomitant Medicat | tions | | |
| 8 | Safety | MH2 | Listing of Medical Conditions | | SAC [1] |
| 9 | Safety | CM3 | Listing of Concomitant Medications | | SAC [1] |
| Expos | ure | | | <u> </u> | |
| 10 | Safety | SAFE_L1 | Listing of Exposure Data | | SAC [1] |
| Safety | | | | | |
| 11 | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC [1] |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 12 | Safety | AE8 | Listing of All Adverse Events | | SAC [1] |
| 13 | Safety | AE8 | Listing of Drug-Related Adverse Events | | SAC [1] |
| 14 | Safety | SAFE_L2 | Listing of Serious Adverse Events | | SAC [1] |
| 15 | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study | | SAC [1] |
| 16 | Safety | SAFE_L3 | Listing of Infusion Site Reaction Adverse Events | Conditional display | SAC [1] |
| 17 | Safety | SAFE_L4 | Listing of Liver Adverse Events | Conditional display | SAC [1] |
| 18 | Safety | SAFE_L5 | Listing of Cardiovascular Adverse Events | Conditional display | SAC [1] |
| 19 | Safety | SAFE_L8 | Listing of Rash Events | Conditional display | SAC [1] |
| Labor | atory Measureme | nts | | | |
| 20 | Safety | LB5 | Listing of Clinical Chemistry Toxicities of Grade 3 or Higher | | SAC [1] |
| 21 | Safety | LB5 | Listing of All Clinical Chemistry Data for Subjects with Toxicities of Grade 3 or Higher | | SAC [1] |
| 22 | Safety | LB5 | Listing of Haematology Toxicities of Grade 3 or Higher | | SAC [1] |
| 23 | Safety | LB5 | Listing of All Haematology Data for Subjects with Toxicities of Grade 3 or Higher | | SAC [1] |
| 24 | Safety | UR2a | Listing of Urinalysis Toxicities of Grade 3 or Higher | | SAC [1] |
| 25 | Safety | UR2a | Listing of Urinalysis Data for Subjects with Toxicities of Grade 3 or Higher | | SAC [1] |
| ECGs | | | · | | |
| 26 | Safety | EG5 | Listing of Abnormal ECG Findings | | SAC [1] |
| 27 | Safety | EG5 | Listing of All ECG Findings for Subjects with an Abnormal Finding | | SAC [1] |
| 28 | Safety | EG3 | Listing of ECG Values of Potential Clinical Importance | | SAC [1] |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 29 | Safety | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC [1] |
| Vital S | Signs | • | | | |
| 30 | Safety | VS4 | Listing of Vital Signs of Potential Clinical Importance | | SAC [1] |
| 31 | Safety | VS4 | Listing of All Vital Signs for Subjects with Potential Clinical Importance Values | | SAC [1] |
| Liver | Events | | | | |
| 32 | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | Conditional display | SAC [1] |
| 33 | Safety | MH3 | Listing of Medical Conditions for Subjects with Liver Stopping Events | Conditional display | SAC [1] |
| 34 | Safety | SAFE_L9 | Listing of Alcohol Intake at Onset of Liver Event | Conditional display | SAC [1] |
| 35 | Safety | PKCL1X | Listing of Plasma Concentration Data for Subjects with Liver Stopping Events | Conditional display | SAC [1] |
| 36 | Safety | LIVER7 | Listing of Liver Biopsy Details | Conditional display | SAC [1] |
| 37 | Safety | LIVER8 | Listing of Liver Imaging Details | Conditional display | SAC [1] |
| Cardia | ac Telemetry | • | | | |
| 38 | Safety | SAFE_L10 | Listing of Cardiac Telemetry Monitoring | | SAC [1] |
| 39 | Safety | SAFE_L11 | Listing of Cytokine Data | | SAC [1] |
| Pharn | nacokinetic Conce | entration | | | |
| 40 | PK | PKCL1X | Listing of GSK3342830 Pharmacokinetic Plasma Concentration-Time Data by Treatment in Part 1 and Part 3 | | SAC [1] |
| 41 | PK | PKUL1P | Listing of GSK3342830 Pharmacokinetic Urine Concentration-Time Data by Treatment in Part 1 and Part 3 | | SAC [1] |

| ICH: | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 42 | PK | PKCL1X | Listing of GSK3342830 Pharmacokinetic Plasma Concentration-Time Data by Treatment in Part 2 | | SAC [1] |
| 43 | PK | PKUL1P | Listing of GSK3342830 Pharmacokinetic Urine Concentration-Time Data by Treatment in Part 2 | | SAC [1] |
| Pharn | Pharmacokinetic Parameter | | | | |
| 44 | PK Parameter | PLPL1X | Listing of GSK3342830 Plasma Pharmacokinetic Parameters by Treatment in Part 1 and Part 3 | | SAC [1] |
| 45 | PK Parameter | PLPL1X | Listing of GSK3342830 Urine Pharmacokinetic Parameters by Treatment in Part 1 and Part 3 | | SAC [1] |
| 46 | PK Parameter | PLPL1X | Listing of GSK3342830 Plasma Pharmacokinetic Parameters by Treatment in Part 2 | | SAC [1] |
| 47 | PK Parameter | PLPL1X | Listing of GSK3342830 Urine Pharmacokinetic Parameters by Treatment in Part 2 | | SAC [1] |

Example : SAFE\_F1 Page 1 of n

Protocol: 204847

Population : Safety

Figure 2.1

Part: xx Cytokine Parameter (Unit)

Boxplot of Cytokine Data

Programming notes: Present each cytokine parameter on a separate page for all scheduled visits. Include a separate line for each treatment and use different symbols for each treatment. Include a legend to describe the treatments.

Visit

Example : SAFE\_F2 Page 1 of n

Protocol: 204847

Population : Safety

Figure 2.2 Part: xx

Individual Cytokine Plot
 Subject = xxxxx



Source Data: Listing 39

Programming notes: Present each subject separately (one per page) and then present all cytokine parameters on the same page for that subject. Include a separate line for each parameter and use different symbols for each parameter. Include a legend to describe the parameters and the units.

Present all scheduled results by visit for the x-axis.


Protocol: 204847 Population: PK

Figure 3.01
Mean (SD) GSK3342830 Single Dose Plasma Concentration-Planned Time Plots for Part 1 and Part 3 (Linear and Semi-Log)

Part: Part 1



Note to Programmer: Present Part 1 first, then Part 3. Dashed line represents the LLQ. Present all dose levels by part in the same plots. Add legend for doses at the bottom.

Source Data: Listing 39


Protocol: 204847
Population: PK

# Figure 3.02 Median (range) GSK3342830 Single Dose Plasma Concentration-Planned Time Plots for Part 1 and Part 3 (Linear and Semi-Log)

Note to Programmer: Present Part 1 first, then Part 3. Display dashed line to represent the LLQ. Present all cohort groups in the same plots. Add legend for doses at the bottom.

Planned Relative Time (Hrs)

Note: LLQ = xx units Source Data: Listing 39

Planned Relative Time (Hrs)


Protocol: 204847 Population: PK

Figure 3.03

Mean (SD) GSK3342830 Plasma Concentration-Planned Time Plots for Part 2 (Linear and Semi-Log)

Day: 1



Note to Programmer: Display dashed line to represent the LLQ. Present all cohort groups in the same plots. Add legend for doses at the bottom. Repeat for Day 15.

Note: LLQ = xx units Source Data: Listing 41


Protocol: 204847
Population: PK

Figure 3.04 Median (range) GSK3342830 Plasma Concentration-Planned Time Plots for Part 2 (Linear and Semi-Log) Day : 1

Linear Scale

Semi-Logarithmic Scale

(strium)
(

Note to Programmer: Display dashed line to represent the LLQ. Present all cohort groups in the same plots. Add legend for doses at the bottom. Repeat for Day 15.

Note: LLQ = xx units Source Data: Listing 41


Protocol: 204847
Population: PK

Figure 3.05
Median (range) GSK3342830 Plasma Pre-dose Concentration versus Day for Part 2 (Linear and Semi-Log)



Note to Programmer: Display dashed line to represent the LLQ. Present all cohort groups in the same plots. Add legend for doses at the bottom.

Note: LLQ = xx units Source Data: Listing 41
Page 1 of n Example : PKCF1P

Protocol: 204847 Population : PK

Figure 3.06 Individual GSK3342830 Single Dose Plasma Concentration-Planned Time Plots for Part 1 and Part 3 (Linear and Semi-Log) Subject ID: XXXX

Part: Part 1

Linear Scale

Semi-Logarithmic Scale

Concentration (units) Actual Relative Time (Hrs)

Actual Relative Time (Hrs)

Note to Programmer: Present Part 1 first, then Part 3. Display dashed line to represent the LLQ.

Note: LLQ = xx units Source Data: Listing 39

Example : PKCF1P

Protocol: 204847 Population: PK

Figure 3.07


Individual GSK3342830 Plasma Concentration-Planned Time Plots for Part 2 (Linear and Semi-Log)
Subject ID: XXXX



Note to Programmer: Display dashed line to represent the LLQ. Display Day 1 and Day 15 on the same figure.

Note: LLQ = xx units Source Data: Listing 41


Protocol: 204847

Population : PK Parameter

Figure 3.08 Comparative Plot of Individual GSK3342830 Plasma AUC(0-t) Versus Dose for Part 1 and Part 3



Note to Programmer: Present box plot for all cohort groups in the same plot. Place Part 3 at the right end of the axis, footnote will be added for the Part 3 dose.


Protocol: 204847

Population : PK Parameter

Figure 3.09
Comparative Plot of Individual GSK3342830 Plasma AUC(0-inf) Versus Dose for Part 1 and Part 3



Note to Programmer: Present box plot for all cohort groups in the same plot. Place Part 3 at the right end of the axis, footnote will be added for the Part 3 dose.3


Protocol: 204847

Population : PK Parameter

Figure 3.10

Comparative Plot of Individual GSK3342830 Plasma Cmax Versus Dose for Part 1 and Part 3



Note to Programmer: Present box plot for all cohort groups in the same plot. Place Part 3 at the right end of the axis, footnote will be added for the Part 3 dose.


Protocol: 204847

Population : PK Parameter

Figure 3.11 Comparative Plot of Individual GSK3342830 Plasma Ae Versus Dose for Part 1



Note to Programmer: Present all cohort groups in the same plots.


Protocol: 204847

Population : PK Parameter

Figure 3.12 Comparative Plot of Individual GSK3342830 Plasma AUC(0-t) Versus Dose on Day 1 for Part 2



Note to Programmer: Present all cohort groups in the same plots.


Protocol: 204847

Population : PK Parameter

Figure 3.13 Comparative Plot of Individual GSK3342830 Plasma AUC(0-inf) Versus Dose on Day 1 for Part 2



Note to Programmer: Present all cohort groups in the same plots.


Protocol: 204847

Population : PK Parameter

Figure 3.14 Comparative Plot of Individual GSK3342830 Plasma Cmax Versus Dose on Day 1 for Part 2



Note to Programmer: Present all cohort groups in the same plots.


Protocol: 204847

Population : PK Parameter

Figure 3.15
Comparative Plot of Individual GSK3342830 Plasma Ae Versus Dose on Day 1 for Part 2



Note to Programmer: Present all cohort groups in the same plots.


Protocol: 204847

Population : PK Parameter

Figure 3.16 Comparative Plot of Individual GSK3342830 Plasma AUC(0-tau) Versus Dose on Day 15 for Part 2



Note to Programmer: Present all cohort groups in the same plots.


Protocol: 204847

Population : PK Parameter

Figure 3.17 Comparative Plot of Individual GSK3342830 Plasma Cmax Versus Dose on Day 15 for Part 2



Note to Programmer: Present all cohort groups in the same plots.


Protocol: 204847

Population : PK Parameter



Note to Programmer: Present all cohort groups in the same plots.

Page 1 of n : PK\_F1 Example

Protocol: 204847

Population : PK Parameter

Figure 3.19 AUC(0-t) (µg.h/mL) in Part 1 - Dose Response Curve



Note: The predictive distributions are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term. Source Table: T3.16

Programming notes:

Example : PK\_F1 Page 1 of n

Protocol: 204847

Population : PK Parameter

Figure 3.20

Cmax (µg/mL) in Part 1 - Dose Response Curve

Note: The predictive distributions are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term.

Programming notes: repeat figure 3.19 for Cmax (µg/mL)

Page 1 of n : PK\_F1 Example

Protocol: 204847

Population : PK Parameter

> Figure 3.21  $AUC(0-8) \times 3$  (µg.h/mL) in Part 2 - Dose Response Curve

Note: The predictive distributions are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term.

Source Table: T3.17

Programming notes: repeat figure 3.19 for AUC[0-8]x3 with X-axis only has 3 dose levels: 1000, 2000, 4000 mg

Example : PK\_F1 Page 1 of n

Protocol: 204847

Population : PK Parameter

Figure 3.22

Cmax (µg/mL) in Part 2 - Dose Response Curve

Note: The predictive distributions are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term. Source Table: T3.17

Programming notes: repeat figure 3.19 for Cmax (µg/mL) with X-axis only has 3 dose levels: 1000, 2000, 4000 mg

Example : TA1 Page 1 of n
Protocol : 204847

Population : Randomized

Listing 1

Listing of Randomized and Actual Treatments

Part: xx

| Subject ID. | Cohort | Randomisation<br>Number | Randomization<br>Date | Randomised Treatmen | t Actual Treatment |
|---|---|---|---|---|---|
| xxx | x | xxxxx | DDMMMYYYY | xxxxxxxxxxx | xxxxxxxxxxx |
| xxx | х | xxxxx | DDMMMYYYY | xxxxxxxxxxx | xxxxxxxxxxx |

Example : ES2
Protocol : 204847

Protocol : 20484/
Population : Safety

Listing 2

Listing of Reasons for Study Withdrawal

Part: xx

| Subject ID. | Date of Withdrawal | Study Day | Primary Reason |
|-------------|--------------------|-----------|----------------|
| xxx | DDMMMYYYY | Х | xxxxxxxxxxx |
| xxx | DDMMMYYYY | х | xxxxxxxxxxxxx |
| xxx | DDMMMYYYY | х | xxxxxxxxxxx |
| xxx | DDMMMYYYY | Х | xxxxxxxxxxxxx |


Example : ES7
Protocol : 204847
Population : Screened

# Listing 3 Listing of Reasons for Screening Failure

| Subject ID. | Date of Screen Failure | Reason |
|-------------|------------------------|---------------|
| xxx | DDMMMYYYY | xxxxxxxxxxx |
| xxx | DDMMMYYYY | xxxxxxxxxxxxx |
| xxx | DDMMMYYYY | xxxxxxxxxxx |
| xxx | DDMMMYYYY | xxxxxxxxxxxxx |

Example : DV2 Page 1 of n

Protocol : 204847
Population : Screened

Listing 4 Listing of Important Protocol Deviations

Part: xx

Treatment: xxxx

Date of Category/ Subject Deviation/ Description ID. Study day Subcategory Outcome xxxxxx/ ddmmmyyyy/ xxxxxxxxxx/ XXXXXXXXXXXXXXXXXXXXXX XXXXXXXX xxxxxx XXXXXXXXX ddmmmyyyy/ xxxxxxxxxx/ xxxxxxxxxxxxx xxxxxxx XX XXXXXXXXX ddmmmyyyy/ xxxxxx/ xxxxxxxxxxxxxxx XXXXXXXXXXXX XXXXXXX XXXXXX xxxxxx/ ddmmmyyyy/ xxxxxxxxxx/ XXXXXXXXXXXX XXXXXXXX XXXXXX XXXXXXXXX

Example : IE3 Page 1 of n Protocol : 204847

Protocol : 204847
Population : Safety

Listing 5

Listing of Subjects with Inclusion/Exclusion Criteria Deviations

Part: xx

| Subject ID. | Туре | Criterion |
|-------------|-----------|---------------|
| xxx | Inclusion | xxxxxxxxxxx |
| XXX | Exclusion | xxxxxxxxxxxx |
| xxx | xxxxxxxxx | xxxxxxxxxxx |
| xxx | xxxxxxxxx | xxxxxxxxxxxxx |


Example : DM2
Protocol : 204847
Population : Safety

Listing 6

Listing of Demographic Characteristics

Part: xx

Treatment: xxxx

| Subject | Year | Age | | | Height | Weight | BMI | _ | Subject Consume | Subject Consume Caffeine/Avg. | Subjects<br>History<br>of Drug |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ID. | Birth | (yrs) | Sex | Ethnicity | (cm) | (kg) | (kg/m^2) | Last Smoked | Consumed Weekly | Servings per Day | Use |
| XXXX | YYYY | xx | Female | Hispanic/Latino | xxx.x | xxx.x | xxx.x | Yes | xx | xx | xx |
| xxxx | YYYY | XX | Female | Not<br>Hispanic/Latino | XXX.X | xxx.x | xxx.x | Yes | xx/DDMMYYYY | xxx/xx | XX |

...

Example : DM9 Page 1 of n Protocol : 204847

Protocol : 20484/
Population : Safety

Listing 7 Listing of Race

Part: xx

Treatment: xxxx

Subject

ID. Race

Example : MH2

Population : Randomized

Listing 8

Listing of Medical Conditions

Part: xx

Treatment: xxxx

Subject Classification PPD - This section has been excluded to protect patient privacy. Condition Status

Example : CM3

Population : Randomized

Listing 9

Listing of Concomitant Medications

Part: xx

| _ Subj. ID | ATC Level 1/<br>Ingredient/<br>Verbatim Text/<br>Indication | Dose/<br>Units/<br>Freq/<br>Route | Start<br>Date/Time<br>Study Day/<br>Period Day | Stop Date/Time<br>Study Day/<br>Period Day | Started<br>Pre-<br>Trial? | Ongoing<br>Medi-<br>cation? |
|---|---|---|---|---|---|---|
| XXXX | <pre>Endocrine &amp; metabolic/ Fluticasone propionate/ FLIXOTIDE/ Asthma</pre> | 2/<br>MG/<br>2XD/<br>IH | 27SEP1999/<br>12:30/<br>15/ | | | Y |

Example : SAFE\_L1 Protocol : 204847 Page 1 of n

Population : Safety

Listing 10 Listing of Exposure Data

Part: xx

| Subject ID. | Treatment | | End<br>Date/Time<br>of Dose | Dose | Dose<br>Unit | Was infusion interrupted?/ Reason/ Interrupt Date/Time/ Restart Date/Time | Was infusion discontinued?/ Reason/ Discontinuation Date/Time | Did subject receive correct treatment?/ |
|---|---|---|---|---|---|---|---|---|
| xxx | XXXXXX | DDMMMYYYY/<br>hh:mm | DDMMMYYYY/<br>hh:mm | XX | xx | No | No | Yes |
| | XXXXXX | DDMMMYYYY/<br>hh:mm | DDMMMYYYY/<br>hh:mm | XX | XX | Yes/xxxxxxxxxx<br>DDMMMYYYY/hh:mm/<br>DDMMMYYYY/hh:mm | Yes/xxxxxxxx<br>DDMMMYYYY/hh:mm | No/xxxxxxxx |

Example : AE7
Protocol : 204847

Protocol : 20484/
Population : Safety

Listing 11

Listing of Subject Numbers for Individual Adverse Events

Part: xx

| System Organ Class | | | |
|--------------------|--------|----------------|----------------------|
| Preferred Term | Group | No. with Event | Subject Numbers |
| SOC #1 | | | |
| Preferred Term #1 | XXXXXX | X | XXXX, XXXXX, XXXXXXX |
| | xxxxxx | X | xxxx, xxxxx, xxxxxxx |
| | | | xxxx, xxxxx, xxxxxxx |
| Preferred Term #2 | xxxxxx | X | xxxx, xxxxx, xxxxxxx |
| | xxxxxx | X | xxxx, xxxxx, xxxxxxx |
| | | | xxxx, xxxxx, xxxxxxx |

Example : AE8
Protocol : 204847
Protocol : 204847

Population : Safety

Listing 12 Listing of All Adverse Events

Part: x

| Subj.<br>ID | Age(y)/<br>Sex/<br>Race/<br>Weight<br>(kg) | System Organ Class/<br>Preferred Term/<br>VERBATIM TEXT | Outcome/ Onset Date/Time Date/Time of Resolution/ Duration | Time Since<br>1st Dose/<br>Time Since<br>Last Dose | Maximum Intensity/ Maximum Serious/ Withdrawal | Frequency/<br>Action Taken/<br>Relation to<br>Study Drug |
|---|---|---|---|---|---|---|
| xxxxx | xx/<br>xxxx/xxx/<br>xx.x | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Resolved/ DDMMMYYYY/hh:mm DDMMMYYYY/hh:mm 1 d | 19 d/<br>19 d/<br>1 d | Mild/<br>No/<br>No | xxxxxxx/<br>Dose reduced/<br>No |
| | | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | Resolving/ DDMMMYYYY/hh:mm DDMMMYYYY/hh:mm 1 d | 21 d/<br>1 d/<br>1 d | Moderate/<br>No/<br>No | xxxxxxx/ Dose inter- rupted/ No |
| | | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | Not resolved/ DDMMMYYYY/hh:mm DDMMMYYYY/hh:mm 120 d | 36 d/<br>16 d/<br>16 d | Severe/<br>No/<br>Yes | xxxxxxx/<br>Withdrawn/<br>No |
| | | xxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxxxxxxxx | Resolved with sequelae/ DDMMMYYYY/hh:mm DDMMMYYYY/hh:mm 85 d | 99 d/<br>79 d/<br>1 d | Mild/<br>No/<br>No | xxxxxxx/<br>None/<br>Possible |


Example : AE8
Protocol : 204847
Population : Safety

Listing 13

Listing of Drug-Related Adverse Events

Note to programmer: Use the same shell as Listing 12.

Protocol : 204847

Population : Safety

Listing 14 Listing of Serious Adverse Events

Part: x

Treatment: xxxxx

Outcome: xxxxxxxxxxxxxxxx

| Subj. | Age(y)/<br>Sex/<br>Race/<br>Weight<br>(kg) | System Organ Class/<br>Preferred Term/<br>VERBATIM TEXT | Onset Date/Time Date/Time of Resolution/ Duration | Time Since<br>1st Dose/<br>Time Since<br>Last Dose | Maximum<br>Intensity/<br>Maximum<br>Serious/<br>Withdrawal | Frequency/<br>Action Taken/<br>Relation to<br>Study Drug |
|---|---|---|---|---|---|---|
| xxxxx | xx/<br>xxxx/xxx/<br>xx.x | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxxxxxxxxx | DDMMMYYYY/hh:mm DDMMMYYYY/hh:mm 1 d | 19 d/<br>19 d/<br>1 d | Mild/<br>No/<br>No | xxxxxxx/<br>Dose reduced/<br>No |
| | | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | DDMMMYYYY/hh:mm DDMMMYYYYY/hh:mm 1 d | 21 d/<br>1 d/<br>1 d | Moderate/<br>No/<br>No | xxxxxxx/ Dose inter- rupted/ No |
| | | ************/ **************/ ********* | DDMMMYYYY/hh:mm<br>DDMMMYYYY/hh:mm<br>120 d | 36 d/<br>16 d/<br>16 d | Severe/<br>No/<br>Yes | xxxxxxx/<br>Withdrawn/<br>No |
| | | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | DDMMMYYYY/hh:mm<br>DDMMMYYYY/hh:mm<br>85 d | 99 d/<br>79 d/<br>1 d | Mild/<br>No/<br>No | xxxxxxx/<br>None/<br>Possible |

## Listing 14 Listing of Serious Adverse Events

Part: x

Treatment: xxxxx

Outcome: xxxxxxxxxxxxxxx

| Subj.<br>ID | Age(y)/<br>Sex/<br>Race/<br>Weight<br>(kg) | System Organ Class/<br>Preferred Term/<br>VERBATIM TEXT | Reason<br>Considered<br>SAE/Recur After<br>Invetigational<br>Product<br>Administered? | Possible<br>Causes of<br>SAE | Relevant<br>Medical<br>Conditions/Onset<br>Date/Present at<br>Time of SAE | Relevant Risk<br>Factors |
|---|---|---|---|---|---|---|
| xxxxx | xx/<br>xxxx/xxx/<br>xx.x | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxx/xx | xxxx:<br>xxxxxxxx | xxxxxxxxxxx<br>(DDMMMYYYY)xxx/ | xxxxx |
| | | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | xxxxxxxxxx/xx | xxxx:<br>xxxxxxxx | xxxxxxxxxxx<br>(DDMMMYYYY)xxx/ | xxxxxxxxxxx |
| | | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | xxxxxxxxxx/xx | xxxx:<br>xxxxxxxx | XXXXXXXXXXX<br>(DDMMMYYYY)XXX/ | |
| | | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxx/<br>xxxxxxxxx | xxxxxxxxxx/xx | xxxx:<br>xxxxxxxx | xxxxxxxxxxx<br>(DDMMMYYYY)xxx/ | xxxxxxx |

#### Listing 14 Listing of Serious Adverse Events

Part: x

Treatment: xxxxx

Outcome: xxxxxxxxxxxxxxx

Relevant Concomitant

Age(y)/ Medications/

Sex/ Dose/Frequency/Route/Taken Prior Subj. Race/ System Organ Class/ Details of to Study/ ΙD Weight Preferred Term/ Start Date/Stop Date/Ongoing/ Investigational Relevant Narrative (kg) VERBATIM TEXT Product Assessments Remarks xxxxx xx/ xxxxxxxxxxxxxx/ xxxxxxxxxxx/xxx (unit)/xxxxx/ XXXXXXXXX XXXXXXXXX XXXXXXXXX xxxx/xxx/ xxxxxxxxxxxxxx/ xxxxxxx/xxx/ DDMMMYYYY/DDMMMYYY/ XX.X xxxxxxxxxxxx XXXXXXXX xxxxxxxxxxxxx/ xxxxxxxxxxx/xxx (unit)/xxxxx/ XXXXXXXXX XXXXXXXXX XXXXXXXXX xxxxxxxxxxxxx/ xxxxxxx/xxx/ xxxxxxxxxxxx DDMMMYYYY/Ongoing/ XXXXXXXX xxxxxxxxxxxxxx/ XXXXXXXXX XXXXXXXXX XXXXXXXXX xxxxxxxxxxxxxx/

XXXXXXXXX

XXXXXXXXX

XXXXXXXXX

XXXXXXXXXXXX

xxxxxxxxxxxxxx/


Example : AE8
Protocol : 204847
Population : Safety

Listing 15

Listing of Adverse Events Leading to Withdrawal from Study

Note to programmer: Use the same shell as Listing 11.

Protocol : 204847

Protocol : 20484/
Population : Safety

Listing 16

Listing of Infusion Site Reaction Adverse Events

Part: xx

| | | | /-! | Reaction<br>Details/ | Reaction<br>Time/ | Require<br>Management?/<br>Photographs | Biopsy<br>Taken?/<br>Interp- | Recent exposure?/ Allergic Reactions Other Drugs?/ |
|---|---|---|---|---|---|---|---|---|
| | | | Date/Time | Skin | Inter- | Taken? | retation/ | History of |
| Subject | AE/SAE | Date of | of | Rash | vention/ | Reaction | Diagnostic | Allergic |
| ID. | Number | Infusion | Reaction | Type | Treatment? | Length, Width (cm) | Tests | Reaction/ |
| xxx | xxxxx | DDMMMYYYY | DDMMMYYYY/<br>hh:mm | xxxxx/<br>xxxxx | xxxxx/<br>xxxxx | xx/<br>xx/<br>xx, xx cm | xx/<br>xxxxxxx/<br>xxxxxxxx | xx/<br>xx/<br>NONE |

Protocol : 204847

Protocol : 204847
Population : Safety

Listing 17

Listing of Liver Adverse Events

Note to programmer: Use the same shell as Listing 11. Present all applicable variables recorded on the eCRF.
Protocol : 204847

Protocol : 204847 Population : Safety

Listing 18

Listing of Cardiovascular Adverse Events

Note to programmer: Use the same shell as Listing 15. Present all applicable variables recorded on the eCRF.

Protocol : 204847

Population : Safety

Listing 19 Listing of Rash Events

Part: xx

Treatment: xxxx

| Subject<br>ID. | Rash Onset<br>Date/Time | Rash Symptoms/<br>Type | Description/ Appearance/ Appearance/ Site | Require Management?/ Photographs Taken? Reaction Length, Width (cm) | Biopsy Taken?/ Interp- retation/ Diagnostic Tests | Recent exposure?/ Allergic Reactions Other Drugs?/ History of Allergic Reaction/ |
|---|---|---|---|---|---|---|
| xxx | DDMMMYYYY/hh:mm | xxxxxxxx/<br>xxxxxxxxxxx | xxxxxxx/<br>xxxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxx | xx/<br>xx/<br>xx, xx cm | xx/<br>xxxxxxx/<br>xxxxxxxx | xx/<br>xx/<br>NONE |

Example : LB5

Population : Safety

Listing 20

Listing of Clinical Chemistry Toxicities of Grade 3 or Higher

Part: xx

Treatment: xxxx

| Subj. | Age(y)/<br>Sex/ | Lab test | Planned | | Study | ( | Converted Data | Flá | ag[1] | |
|---|---|---|---|---|---|---|---|---|---|---|
| ID | Race | (units) | Relative Time | Date | Day | Value | Normal Range | NR | TG | BL |
| xxxxx | xx/<br>xxxx/<br>xxxxxx | xxxxxx (xxx) | xxxxxx | DDMMMYYYY<br>DDMMMYYYY | x<br>x | xx.x<br>xx.x | xx.x-xx.x<br>xx.x-xx.x | | | |
| [1] ND | fan Namal | XXXXXX (XXX) | XXXXXXXX<br>XXXXXXXX | DDMMMYYYY<br>DDMMMYYYY | X<br>X | XX.X<br>XX.X | XX.X-XX.X<br>XX.X-XX.X | H<br>I-Rolow r | Х | Н |

<sup>[1]</sup> NR for Normal Range flag, TG for Toxicity flag; BL for Change from Baseline flag. H=Above range, L=Below range

Example : LB5
Protocol : 204847
Population : Safety

Listing 21

Listing of All Clinical Chemistry Data for Subjects with Toxicities of Grade 3 or Higher

Note to programmer: Use the shell from Listing 20.

Example : LB5
Protocol : 204847
Population : Safety

Listing 22

Listing of Haematology Toxicities of Grade 3 or Higher

Note to programmer: Use the shell from Listing 20.

Example : LB5
Protocol : 204847
Population : Safety

Listing 23

Listing of Haematology Data for Subjects with Toxicities of Grade 3 or Higher

Note to programmer: Use the shell from Listing 20.

Example : UR2a Page 1 of n Protocol : 204847

Protocol : 204847
Population : Safety

Listing 24

Listing of Urinalysis Toxicities of Grade 3 or Higher

Part: xx

Treatment: xxxx

| Subject ID. | Visit | Sample Date | Sample Time | Study Day | Urinalysis Test | Result | Toxicity<br>Grade |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxx | DDMMMYYYY | HH:MM | 1 | Blood | ++ or 2+ | Х |
| | XXXXX | DDMMMYYYY | HH:MM | 1 | Blood | + or 1+ | |
| xxxxxx | xxxxx | DDMMMYYYY | HH:MM | 1 | Blood | + or 1+ | |
| | | | | | Protein | +++ or 3+ | x |
| | XXXXX | DDMMMYYYY | HH:MM | 1 | Blood | + or 1+ | |

Example : UR2a Page 1 of n

Example : UR2a Protocol : 204847 Population : Safety

Listing 25

Listing of Urinalysis for Subjects with Toxicities of Grade 3 or Higher

Note to programmer: Use the shell from Listing 24.

Example : EG5

Population : Safety

Listing 26

Listing of Abnormal ECG Findings

Part: xx

| Part: x | | | | | | |
|---|---|---|---|---|---|---|
| Treatme<br>Subj. | Age/<br>Sex/<br>Race | Planned Rel<br>Time/<br>ECG Date/<br>Time | Study<br>Day | ECG Finding | Clinically<br>Significant<br>Change from<br>Baseline? | Clinically<br>Significant Abnormality |
| xxxxx | xx/<br>xxxxx/<br>xxxx | xxxxxxx/<br>DDMMMYYYY<br>/hh:mm | xx | Abnormal-not<br>clinically<br>significant | No | |
| | | xxxxxxx/<br>DDMMMYYYY<br>/hh:mm | XX | Abnormal-not<br>clinically<br>significant | No | |
| | | xxxxxxx/<br>DDMMMYYYY<br>/hh:mm | xx | Abnormal-clinically significant | Yes | Sinus tachycardia |
| | | xxxxxxx/<br>DDMMMYYYY<br>/hh:mm | XX | Abnormal-not<br>clinically<br>significant | No | |
| xxxxx | xx/<br>xxxxx/<br>xxxx | xxxxxx/<br>DDMMMYYYY<br>/hh:mm | XX | Abnormal-clinically significant | Yes | Ectopic ventricular beats |
| | | xxxxxx/<br>DDMMMYYYY<br>/hh:mm | XX | Abnormal-clinically significant | No | Ectopic ventricular beats |

Example : EG5
Protocol : 204847
Population : Safety

Listing 27

Listing of All ECG Findings for Subjects with an Abnormal Finding

Note to programmer: Use the shell from Listing 26.

Example : EG3
Protocol : 204847

Population : Safety

Listing 28

Listing of ECG Values of Potential Clinical Importance

Part: xx

Treatment: xxxx

| | Age/ | | | | Heart<br>Rate | PR<br>Inter- | QRS<br>Dura- | QRS | QT<br>Inter- | QTc<br>Inter- | QTc<br>(Baz- | QTc<br>(Frid- | RR<br>Inter- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subj. ID | Sex/ | Planned | | Study | | val | tion | Axis | val | val | ett) | ericia) | val |
| 5 - | Race | Rel Time | ECG Date/ Time | Day | min.) | (msec) | (msec) | (deg) | (msec) | (msec) | (msec) | (msec) | (msec) |
| XXXXXX | xx/<br>xxxxxx/ | XXXXXX | DDMMMYYYY/hh:mm | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | XXXXX | | | | | | | | | | | | |
| | | XXXXXXX | DDMMMYYYY/hh:mm | XX | XX | xx L | XX | XX | XX | XX | XX | XX | XX |
| | | XXXXXXX | DDMMMYYYY/hh:mm | XX | 80 | XX | XX | XX | XX | XX | XX | XX | XX |
| | | XXXXXXX | DDMMMYYYY/hh:mm | XX | XX | XX | XX | XX | XX | xx H | XX | XX | XX |
| XXXXX | xx/ | XXXXXXX | DDMMMYYYY/hh:mm | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | xxxxxx/ | | | | | | | | | | | | |
| | XXXXX | | | | | | | | | | | | |
| | | XXXXXXX | DDMMMYYYY/hh:mm | XX | XX | XX | XX | XX | XX | xx I | XX | XX | XX |

Note: L=Low, H=High, I=Increase, D=Decrease

Example : EG3 Page 1 of n

Example : EG3
Protocol : 204847
Population : Safety

Listing 29

Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance

Note to programmer: Use shell for Listing 28.

Protocol : 204847

Population : Safety

Listing 30

Listing of Vital Signs of Potential Clinical Importance

Part: xx

Treatment: xxxx

| Subj. ID | Age(y)/<br>Sex/<br>Race | Planned<br>Relative<br>Time | Actual<br>Date/Time | Body<br>Position | Study<br>Day | Systolic<br>Blood<br>Pressure<br>(mmHg) | Diastolic<br>Blood<br>Pressure<br>(mmHg) | Pulse<br>(beats/<br>min) | Temper-<br>ature<br>(C) | Comment |
|---|---|---|---|---|---|---|---|---|---|---|
| xxx | xx/<br>xxxxxx/<br>xxxxx | xxxxxx | DDMMMYYYY/hh:mm | XXXXXXX | Х | xxx | xxx | XXX | XXX | |
| | | xxxxxx | DDMMMYYYY/hh:mm | xxxxxx | Х | XXX | XXX | xxx | | |
| | | xxxxxx | DDMMMYYYY/hh:mm | xxxxxx | Х | Xxx H | Xxx H | xxx | | xxxxxxxxx |
| | | XXXXXXX | DDMMMYYYY/hh:mm | XXXXXX | X | XXX | XXX | XXX | | |
| | | XXXXXXX | DDMMMYYYY/hh:mm | XXXXXX | X | XXX | XXX | XXX | | |
| | | XXXXXXX | DDMMMYYYY/hh:mm | XXXXXX | X | XXX | XXX | XXX | | |
| | | XXXXXXX | DDMMMYYYY/hh:mm | XXXXXXX | X | XXX | XXX | xxx L | | |
| XXX | xx/ | XXXXXXX | DDMMMYYYY/hh:mm | XXXXXXX | X | XXX | XXX | XXX | XXX | |
| | xxxxxx/<br>xxxxx | | | | | | | | | |
| | | XXXXXXX | DDMMMYYYY/hh:mm | xxxxxx | Х | XXX | XXX | xxx | | |

Note: L=Low, H=High


Example : VS4
Protocol : 204847
Population : Safety

Listing 31

Listing of All Vital Signs for Subjects with Potential Clinical Importance Values

Note to programmer: Use shell for Listing 30.

Protocol : 204847
Population : Safety

Listing 32

Listing of Liver Monitoring/Stopping Event Reporting

Part: xxxxx

Treatment: xxxxxx

Time Time

Since Since Restart/Re-challenge

Site Id./ Age (YEARS) / Date First First Last After Stopping

Unique Subject Id. Sex/ Maximum Status of the Detected/ Dose Dose Criteria Was Met Resolved?/
Race Detail Liver Event Study Day (days) (days) Date resolved

PPD - This section has been excluded to protect patient privacy.

Example: MH2 Page 1 of n

Example : MH2
Protocol : 204847
Population : Safety

Listing 33

Listing of Medical Conditions for Subjects with Liver Stopping Events

Part: xx

Treatment: xxxx

| Subject ID | Classification | Condition | Status |
|---|---|---|---|
| xxxx | xxxxxxxxxx<br>xxxxxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Current<br>Past |
| XXXX | xxxx | xxxxxxxxxxxxxx | Current |
| xxxx | xxxxxxxxxx | xxxxxxxxxxxxxxxx | Current |

Example : SAFE\_L9
Protocol : 204847


Protocol : 204847
Population : Safety

Listing 34

Listing of Alcohol Intake at Onset of Liver Event

Part: xx

Treatment: xxxx

Age(y)/

Sex/

| Subject ID | Race | Exam Date/Time | Consume Alcohol? | Average Number Units Consumed per Week? |
|---|---|---|---|---|
| xxxx | xx/xx/xxxxxx | DDMMMYYYY/hh:mm | xxx | х |
| xxxx | xx/xx/xxxxxx | DDMMMYYYY/hh:mm | xx | xx |
| XXXX | xx/xx/xxxxxxx | DDMMMYYYY/hh:mm | XX | X |

Example : PKCL1X
Protocol : 204847

Protocol : 204847 Population : Safety

Listing 35

Listing of Plasma Concentration Data for Subjects with Liver Stopping Events

Note to programmer: Use shell for Listing 40.

Example : LIVER7
Protocol : 204847

Protocol : 204847 Population : Safety

Listing 36
Listing of Liver Biopsy Details

Part: xx

Treatment: xxxx

Age(y)/

| Subject<br>ID | Sex/<br>Race | Biopsy Date/<br>Study Day | Biopsy Size | Liver Biopsy Test | Liver Biopsy Result |
|---|---|---|---|---|---|
| XXXX | xx/<br>xxxxxx/<br>xxxxx | DDMMMYYYY/<br>xx | xx | xxxxxxxxxxx | xxxxxxxxxxxxxxxxx |
| | | | | xxxxxxxxxxx | xxxxxxxxxxxxxxxxxx |
| | | | | xxxxxxxxxxxx | xxxxxxxxxxxxxxxxxx |
| | | | | xxxxxxxxxxx | xxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXXXXXXX | xxxxxxxxxxxxxxxxxx |

Example : LIVER8
Protocol : 204847

Protocol : 204847 Population : Safety

ropulation . Salety

Listing 37

Listing of Liver Imaging Details

Part: xx

Treatment: xxxx

| Subject<br>ID | Age(y)/<br>Sex/<br>Race | Imaging Date/<br>Study Day | Liver Imaging<br>Method | Are Images<br>Technically<br>Adequate | Liver Imaging Test | Liver Imaging Result |
|---|---|---|---|---|---|---|
| xxxx | xx/<br>xxxxxx/ | DDMMMYYYY/<br>xx | xx | xxxx | xxxxxxxxxxx | xxxxxxxxxxxxxxxx |
| | XXXXX | | | | xxxxxxxxxxx | xxxxxxxxxxxxxxx |
| | | | | | XXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXX |
| | | | | | XXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXX |
| | | | | | xxxxxxxxxxx | XXXXXXXXXXXXXXXXXXXXX |

Example : SAFE\_L10 Page 1 of n Protocol : 204847

Protocol : 204847
Population : Safety

Listing 38

DDMMMYYYY/hh:mm DDMMMYYYY/hh:mm xxxxxxxxxxx

Listing of Cardiac Telemetry Monitoring

Part: xx

XXXX

Treatment: xxxx

| Subject ID | Start Date/Time | End Date/Time | Overall Interpretation | Specify Abnormality/Comments |
|---|---|---|---|---|
| xxxx | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm | xxxxxxxxxx | xxxxxxxxxx/xxxxxx |
| xxxx | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm | xxxxxxxx | |

Example : LB5
Protocol : 204847
Population : Safety

Listing 39 Listing of Cytokine Data

Note to programmer: Use the shell from Listing 20. Do not present toxicity (TG) column.

Population : PK

## Listing 40

Listing of GSK3342830 Pharmacokinetic Plasma Concentration-Time Data by Treatment in Part 1 and Part 3

Part: Part 1
Dose: XXXX mg

| Dose: XX | XX mg | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID. | Age (y)/ Sex/ Race xx/ xxxx/ | Visit | Date | Study Day | Planned<br>Relative<br>Time | Actual Time | Time<br>Deviation<br>(h) | Actual Relative<br>Time (h) | Concentration (units) |
| xxxx | XXXXX | XXXX | MMDDYYYY | 1 | pre-dose | HH:MM | XX | 0h 0m 0s | xx.xx |
| | | | | | 0.5h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 1h | HH:MM | XX | 0h 0m 0s | xx.xx |
| | | | | | 1.25h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 1.5h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 2h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 3h | HH:MM | XX | 0h 0m 0s | xx.xx |
| | | | | | 3.5h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 4h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 4.5h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 5h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 6h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 8h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 10h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 12h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 16h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | 2 | 24h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 36h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | 3 | 48h | HH:MM | XX | 0h 0m 0s | XX.XX |

Note to Programmer: Present all Part 1 first, then repeat for Part 3. Please list all the concentration data including unscheduled.

LLOQ = xx.x (units)

NQ=Not quantifiable

Population : PK

Listing 41

Listing of GSK3342830 Pharmacokinetic Urine Concentration-Time Data by Treatment in Part 1 and Part 3

Part: Part 1

| Total Actual Urine Sample |
|---------------------------|
| - |
| of Dunation Cons. Walsons |
| of Duration Conc. Volume |
| ion (h) (units) (units) |
| HH MM xx.xx xx.xx |
| HH MM xx.xx xx.xx |
| HH MM xx.xx xx.xx |
| HH MM xx.xx xx.xx |
| HH MM xx.xx xx.xx |

Note to Programmer: Present all Part 1 first, then repeat for Part 3. Please list all the concentration data including unscheduled.

LLOQ = xx.x (units)

NQ=Not quantifiable

Population : PK

Listing 42
Listing of GSK3342830 Pharmacokinetic Plasma Concentration-Time Data by Treatment in Part 2

| Dose: XX | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Age<br>(y)/<br>Sex/ | | 5. | | Planned<br>Relative | 2 | Time<br>Deviation | Actual Relative | Concentration |
| D. | Race<br>xx/<br>xxxx/ | Visit | Date | Study Day | Time | Actual Time | (h) | Time (h) | (units) |
| XXX | XXXXX | XXXX | MMDDYYYY | 1 | pre-dose | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 0.5h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 1h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 1.25h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 1.5h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 2h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 16h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | 2 | 24h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | 3 | pre-dose | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | 6 | pre-dose | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | 9 | pre-dose | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | 12 | pre-dose | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | 13 | pre-dose | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | 15 | pre-dose | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 0.5h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 1h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 1.25h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 6h | HH:MM | XX | 0h 0m 0s | XX.XX |
| | | | | | 8h | HH:MM | XX | 0h 0m 0s | XX.XX |

Note to Programmer: Please list all the concentration data including unscheduled. Timepoints on day 1 is Pre-dose, 0.5, 1.25,1.5, 2,2.5,3,3.5,4,4.5,5,6,8,10,12,16 and 24. Timepoints on day 15 is Pre-dose, 0.5,1,1.25,1.5,2,2.5,3,3.5,4,4.5, 5, 6 and 8.

LLOQ = xx.x (units) NQ=Not quantifiable Example : PKUL1P
Protocol : 204847
Population : PK Page 1 of n

Listing 43 Listing of GSK3342830 Pharmacokinetic Urine Concentration-Time Data by Treatment in Part 2

| Dose: XXX | KX mg | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID. | Age<br>(y)/<br>Sex/<br>Race | Visit | Date | Study<br>Day | Planned<br>Relative<br>Time | Actual<br>Midpt. of<br>Collection | Actual<br>Duration<br>(h) | Urine<br>Conc.<br>(units) | Total<br>Sample<br>Volume<br>(units) |
| XXXX | xx/<br>xxxx/<br>xxxxx | xxxx | MMDDYYYY | 1 | 0-8h | нн мм | нн мм | XX.XX | XX.XX |
| | | | | 15 | 8-24h<br>0-8h<br>8-24h | НН ММ<br>НН ММ<br>НН ММ | HH MM<br>HH MM<br>HH MM | xx.xx<br>xx.xx<br>xx.xx | xx.xx<br>xx.xx<br>xx.xx |

Note to Programmer: Please list all the concentration data including unscheduled.

LLOQ = xx.x (units) NQ=Not quantifiable

Population : PK Parameter

Part: Part 1
Dose: XXX mg

| 2000 | 9 | | | | |
|---------|----------|----------|-----------|---------|--------|
| | Age (y)/ | | | | |
| Subject | Sex/ | AUC(0-t) | AUC (0-∞) | Cmax | Tmax |
| ID. | Race | (units) | (units) | (units) | (unit) |
| XXXX | xx/ | XX.XX | XX.XX | XX.XX | XX.XX |
| | xxxx/ | | | | |
| | XXXXX | | | | |
| XXXX | xx/ | XX.XX | XX.XX | XX.XX | XX.XX |
| | xxxx/ | | | | |
| | XXXXX | | | | |
| XXXX | xx/ | XX.XX | NC | XX.XX | XX.XX |
| | xxxx/ | | | | |
| | XXXXX | | | | |
| XXXX | xx/ | XX.XX | XX.XX | XX.XX | XX.XX |
| | xxxx/ | | | | |
| | XXXXX | | | | |
| | XXXXX | | | | |

Note to Programmer: Present all Part 1 first, then repeat for Part 3
Additional parameters include t1/2, CL, Vss, %AUCex, tlast, lambda\_z, lambda\_z\_lower, lambda\_z\_upper, lambda\_z\_no. of points

Population : PK Parameter

## Listing 45

Listing of GSK3342830 Urine Pharmacokinetic Parameters by Treatment in Part 1 and Part 3

Part: Part 1
Dose: XXX mg

| B000. 111111 | 9 | | | |
|--------------|----------|---------|---------|-----------|
| | Age (y)/ | | | |
| Subject | Sex/ | Ae | CLr | Feu (0-4) |
| ID. | Race | (units) | (units) | (units) |
| XXXX | xx/ | XX.XX | XX.XX | XX.XX |
| | xxxx/ | | | |
| | XXXXX | | | |
| XXXX | xx/ | XX.XX | XX.XX | XX.XX |
| | xxxx/ | | | |
| | XXXXX | | | |
| | , | | | |
| XXXX | xx/ | XX.XX | XX.XX | XX.XX |
| | xxxx/ | | | |
| | XXXXX | | | |
| | / | | | |
| XXXX | xx/ | XX.XX | XX.XX | XX.XX |
| | xxxx/ | | | |
| | XXXXX | | | |

Note to Programmer: Present all Part 1 first, then repeat for Part 3
Additional parameters include Feu(4-8) (units), Feu(8-12) (units), Feu (12-24) (units), Feu (24-48) (units)

Population : PK Parameter

Listing 46
Listing of GSK3342830 Plasma Pharmacokinetic Parameters by Treatment in Part 2

| Dose: XXX | mg | | | | | |
|---|---|---|---|---|---|---|
| Subject | Age (y)/<br>Sex/<br>Race | Day | AUC(0-t)<br>(units) | AUC(0-∞)<br>(units) | AUC(0-τ) (units) | Cmax<br>(unit) |
| XXXX | xx/<br>xxxx/<br>xxxxx | 1 | xx.xx | xx.xx | xx.xx | xx.xx |
| | | 15 | xx.xx | XX.XX | XX.XX | XX.XX |
| XXXX | xx/<br>xxxx/<br>xxxxx | 1 | xx.xx | xx.xx | xx.xx | xx.xx |
| | | 15 | xx.xx | xx.xx | xx.xx | xx.xx |
| XXXX | xx/<br>xxxx/<br>xxxxx | 1 | xx.xx | NC | xx.xx | xx.xx |
| | | 15 | xx.xx | NC | xx.xx | xx.xx |
| XXXX | xx/<br>xxxx/<br>xxxxx | 1 | xx.xx | xx.xx | xx.xx | xx.xx |
| | | 15 | XX.XX | XX.XX | XX.XX | XX.XX |

#### Note to Programmer:

Additional parameters include Tmax, t1/2, CL, Vss, C $\tau$ , Ratio of time invariance, Ratio of accumulation, %AUCex, tlast, lambda\_z\_lower, lambda\_z\_upper, lambda\_z\_no. of points

Population : PK Parameter

Listing 47
Listing of GSK3342830 Urine Pharmacokinetic Parameters by Treatment in Part 2

Dose: XXX mg Age (y)/ Subject Sex/ Аe CLr Feu (0-8) ID. Race (units) (units) (units) Day XXXX xx/ XX.XX XX.XX XX.XX xxxx/ XXXXX 15 xx.xx xx.xx xx.xx xx/ 1 XXXX XX.XX XX.XX XX.XX xxxx/ XXXXX 15 xx.xx xx.xx xx.xx XXXX xx/ 1 XX.XX XX.XX XX.XX xxxx/ XXXXX 15 XX.XX xx.xx xx.xx xx/ 1 XXXX XX.XX XX.XX XX.XX xxxx/ XXXXX 15 XX.XX XX.XX xx.xx

Note to Programmer:

Additional parameters include Feu(8-24) (units).

Example : NS1 Page 1 of n

Protocol : 204847
Population : Safety

Study Part: 1

| Country | Site ID | Investigator<br>Name | GSK3342830 250 mg<br>(N=xx) | GSK3342830 500 mg (N=xx) | <br>Placebo (N=xx) | Total (N=xx) |
|---|---|---|---|---|---|---|
| xxxxxxxxx | xxxxxxxx | xxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxxxxx | xxxxxxxx | xxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note to programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.


Protocol : 204847
Population : Safety

Table 1.2
Summary of Subject Disposition

Study Part: 1

| | | 12830 250 mg GSK3342830 500 mg Placebo (N=xx) (N=xx) | | | Total<br>(N=xx) | | | |
|---|---|---|---|---|---|---|---|---|
| Subject Status | | | | | | | | |
| Completed | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Withdrawn | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Primary reason for study withdrawal | | | | | | | | |
| Adverse Event | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Protocol Deviation | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Subject reached protocol-defined stopping criteria | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Study closed/terminated | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Lost to Follow-up | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Investigator discretion | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Withdrew Consent | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Other | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |

Note to programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.

Protocol : 204847

Protocol : 204847
Population : Screened

# Table 1.3 Summary of Reasons for Screening Failures

| bananary or neasons for ber | cening rarrares |
|-------------------------------------------|-----------------|
| | Screened |
| | Subjects |
| | (N=xx) |
| Screening Status | |
| Enrolled | xx (xx.x%) |
| Failed | xx (xx.x%) |
| Reason for failure | |
| Did not meet inclusion/exclusion criteria | xx (xx.x%) |
| Adverse event | xx (xx.x%) |
| Protocol deviation | xx (xx.x%) |
| Medical or Surgical Condition Exclusion | xx (xx.x%) |
| Investigator discretion | xx (xx.x%) |
| Participant withdrew consent | xx (xx.x%) |
| Lost to follow up | xx (xx.x%) |
| Other | xx (xx.x%) |

Example : DV1

Protocol : 204847
Population : Screened


Table 1.4
Summary of Important Protocol Deviations

Study Part: 1

| Category/Subcategory | GSK3342830 250 mg | GSK3342830 500 mg | <br>Placebo | Total |
|---|---|---|---|---|
| catedot A, princatedot A | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any protocol deviations | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) | xx (xx.x%) |
| Informed Consent | | | | |
| XXXXXXXXXXXX | | | | |
| xxxxxxxxxxx | | | | |
| ••• | | | | |
| Eligibility criteria not met xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) | xx (xx.x%) |
| Not withdrawn after developing withdrawal criteria | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) | xx (xx.x%) |
| Excluded medication, vaccine, or device | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) | xx (xx.x%) |
| Visit Completion | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) | xx (xx.x%) |
| Assessment or time point completion | | | | |
| Wrong study treatment/administration/dose or incorrect dose | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) | xx (xx.x%) |
| Study Procedures | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) | xx (xx.x%) |
| Failure to report safety events per protocol | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) | xx (xx.x%) |

Note to programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages. Present all Categories and Subcategories on the eCRF for which there is non-zero count.

Protocol : 204847

Population : Safety

Table 1.5
Summary of Demographic Characteristics

Study Part: 1

| | | GSK3342830 250 mg GS<br>(N=xx) | K3342830 500 mg<br>(N=xx) | | Total<br>(N=xx) |
|---|---|---|---|---|---|
| Sex | n | XX | XX | | XX |
| 7011 | Male | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) |
| | Female | xx (xx.x%) | xx (xx.x%) | ••• | xx (xx.x%) |
| | remare | AA (AA.A.) | AA (AA.A0) | | AA (AA.A0) |
| Age (YEARS)[1] | n | xx | XX | | XX |
| | Mean | XX.X | XX.X | | XX.X |
| | SD | xx.xx | xx.xx | | XX.XX |
| | Median | xx.x | xx.x | | XX.X |
| | Min. | xx.x | xx.x | | XX.X |
| | Max. | XX.X | XX.X | | XX.X |
| Sthnicity | n | XX | XX | | XX |
| | Hispanic/Latino | xx (xx.x%) | xx (xx.x%) | ••• | xx (xx.x%) |
| | Not Hispanic/Latino | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) |
| | Not hippanie, latino | (222.210) | 7171 (1121 • 21 0 ) | | (2121 • 21 0 ) |
| leight (cm) | n | XX | XX | | XX |
| | Mean | XX.X | XX.X | | XX.X |
| | SD | XX.XX | XX.XX | | XX.XX |
| | Median | XX.X | XX.X | | XX.X |
| | Min. | XX.X | XX.X | | XX.X |
| | Max. | XX.X | XX.X | | XX.X |
| Weight (kg) | n | XX | XX | | XX |
| | Mean | XX.X | XX.X | | XX.X |
| | SD | XX.XX | XX.XX | | XX.XX |
| | Median | XX.X | XX.X | ••• | XX.X |
| | Min. | XX.X | XX.X | | XX.X |
| | Max. | XX.X | XX.X | ••• | XX.X |
| BMI (kg/m2) | n | XX | XX | | XX |
| (119/1112/ | Mean | XX.X | XX.X | | XX.X |
| | SD | XX.XX | XX.XX | | XX.XX |
| | Median | XX.X | XX.X | ••• | XX.X |
| | Min. | | | ••• | |
| | Max. | XX.X | XX.X | ••• | XX.X |
| | Max. | XX.X | XX.X | | XX.X |

<sup>[1]</sup> Age is imputed when full date of birth is not provided.


Protocol : 204847
Population : Safety

Table 1.6

Summary of Age Ranges

Study Part: 1

GSK3342830 250 mg GSK3342830 500 mg Total

(N=xx) (N=xx) ... (N=xx)

Age Ranges [1]

Adult (18-64 years) xx (xx.x%) xx (xx.x%) ... xx (xx.x%)

Note to programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.

[1] Age is imputed when full date of birth is not provided.

Protocol : 204847 Population : Safety

Table 1.7 Summary of Race and Racial Combinations

| | GSK3342830 250 mg | GSK3342830 500 mg | Total |
|---|---|---|---|
| Race | (N=xx) | (N=xx) | (N=xx) |
| n AMERICAN INDIAN OR ALASKA NATIVE ASIAN BLACK OR AFRICAN AMERICAN NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER WHITE MULTIPLE | xx<br>xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Programmer's note: Do not display "MULTIPLE" unless present in the data. Percentages will add up to 100. Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.


Protocol : 204847 Population : Safety

Table 1.8 Summary of Race and Racial Combinations Details

| | | GSK3342830 250 mg GSK3342830 500 mg | | Total |
|---|---|---|---|---|
| | | (N=XX) | (N=xx) | (N=xx) |
| Race n | | XX | XX | XX |
| 1A | MERICAN INDIAN OR ALASKA NATIVE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| AS | SIAN | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ВІ | LACK OR AFRICAN AMERICAN | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| N/ | ATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| WI | HITE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.

Example : MH1 Page 1 of n

Protocol : 204847
Population : Safety

Study Part: 1

| _Classification | GSK3342830 250 mg<br>(N=xx) | GSK3342830 500 mg<br>(N=xx) | | Placebo<br>(N=xx) | Total (N=xx) |
|---|---|---|---|---|---|
| Any condition | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Angina pectoris | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Myocardial infarction | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Stroke | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| • • • | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note to programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.


Protocol : 204847 Population : Safety

 ${\tt Table~2.1} \\ {\tt Relationship~of~Adverse~Event~System~Organ~Classes,~Preferred~Terms~and~Verbatim~Text} \\$ 

| System Organ Class | Preferred Term | Verbatim Text |
|--------------------|--------------------|---------------|
| SOC #1 | Preferred Term # 1 | xxxxxxxx |
| | Preferred Term # 2 | XXXXXXXX |
| | Preferred Term # 3 | XXXXXXXX |
| | Preferred Term # 4 | XXXXXXXX |
| SOC #2 | Preferred Term # 1 | XXXXXXXX |
| | Preferred Term # 2 | XXXXXXXX |
| | Preferred Term # 3 | XXXXXXXX |
| | Preferred Term # 4 | XXXXXXXX |

Example : AE1
Protocol : 204847

Population : Safety


Table 2.2 Summary of All Adverse Events

Study Part: 1

| System Organ Class | GSK3342830 250 mg | GSK3342830 500 mg | Total |
|---|---|---|---|
| Preferred Term | (N=xx) | (N=xx) | <br>(N=xx) |
| Any Event | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| System Organ Class #1 | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| Preferred Term #1 | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| Preferred Term #2 | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| Preferred Term #3 | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |

. . .

Note to programmer: System Organ Class (SOC) is displayed in descending order of frequency for 'Overall' then alphabetically. Preferred Term is displayed in descending order of frequency for 'Overall' then alphabetically within SOC.

Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.

Protocol : 204847

Protocol : 204847
Population : Safety

Table 2.3 Summary of Drug-Related Adverse Events

Study Part: 1

| System Organ Class | GSK3342830 250 mg | GSK3342830 500 mg | Total |
|---|---|---|---|
| Preferred Term | (N=xx) | (N=xx) | <br>(N=xx) |
| Any Event | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| System Organ Class #1 | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| Preferred Term #1 | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| Preferred Term #2 | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| Preferred Term #3 | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |

. . .

Note to programmer: System Organ Class (SOC) is displayed in descending order of frequency for 'Overall' then alphabetically. Preferred Term is displayed in descending order of frequency for 'Overall' then alphabetically within SOC.

Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.


Protocol : 204847
Population : Safety

Table 2.4

Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences)

Study Part: 1

| System Organ Class<br>Preferred Term | | GSK3342830 250 mg<br>(N=xx) | GSK3342830 500 mg<br>(N=xx) | <br>Total<br>(N=xx) |
|---|---|---|---|---|
| Any Event | Number of Subject with AEs | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| | Number of AEs | XX | XX | xx |
| System Organ Class #1 | | | | |
| Preferred Term #1 | Number of Subject with AEs | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| | Number of AEs | XX | XX | xx |

Note to programmer: System Organ Class (SOC) is displayed in descending order of frequency for 'Overall' then alphabetically. Preferred Term is displayed in descending order of frequency for 'Overall' then alphabetically within SOC.

Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.

Example : AE16
Protocol : 204847
Population : Safety


Table 2.5

Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences)

Study Part: 1

| System Organ Class<br>Preferred Term | | GSK3342830 250 mg<br>(N=xx) | GSK3342830 500 mg<br>(N=xx) | <br>Total<br>(N=xx) |
|---|---|---|---|---|
| Any Event | Number of Subjects with SAEs | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| | Number of SAEs | xx | XX | XX |
| | Number of Drug-<br>related SAEs | XX | XX | XX |
| | Number of Fatal SAEs | XX | XX | XX |
| | Number of Drug-<br>related Fatal SAEs | xx | xx | xx |
| System Organ Class #1 | | | | |
| Preferred Term #1 | Number of Subjects<br>with SAEs | xx (xx.x%) | xx (xx.x%) | <br>xx (xx.x%) |
| • • • | Number of SAEs | xx | XX | XX |
| | Number of Drug-<br>related SAEs | XX | XX | XX |
| | Number of Fatal SAEs | XX | XX | XX |
| | Number of Drug-<br>related Fatal SAEs | XX | XX | XX |

Note to programmer: System Organ Class (SOC) is displayed in descending order of frequency for 'Overall' then alphabetically. Preferred Term is displayed in descending order of frequency for 'Overall' then alphabetically within SOC.

Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.

Example : LB1
Protocol : 204847
Population : Safety


Table 2.6
Summary of Clinical Chemistry Values

Study Part: 1

| Lab Test | Treatment | N | Planned Relative Time | n | Mean | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXXXX (XXX) | GSK3342830 250<br>mg | XXX | Baseline | XX | xx.x | XX.XX | xx | XX | XX |
| | | | Day 2 | XX | XX.X | XX.XX | XX | XX | XX |
| | | | Follow-Up | XX | XX.X | XX.XX | XX | XX | XX |
| | GSK3342830 500<br>mg | XXX | Baseline | XX | XX.X | XX.XX | xx | XX | XX |
| | , | | Day 2 | XX | xx.x | XX.XX | XX | xx | xx |
| | | | Follow-Up | XX | XX.X | XX.XX | XX | XX | XX |
| | | XXX | Baseline | XX | XX.X | XX.XX | xx | XX | XX |
| | | | Day 2 | XX | XX.X | XX.XX | XX | XX | XX |
| | | | Follow-Up | XX | XX.X | xx.xx | XX | XX | XX |

Note to programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages. Timepoints for Part 1 and Part 3 are Baseline, Day 2, Follow-Up. Timepoints for Part 2 are Baseline, Day 2, Day 5, Day 10, Day 15, and Follow-Up.

Note: For subjects Baseline is defined as the last nonmissing measurement before dosing.

Unscheduled measurements are not included in this summary table except when calculating baseline.


Protocol : 204847
Population : Safety

Table 2.7

Summary of Clinical Chemistry Change from Baseline

Note to programmer: Please use the shell from Table 2.6 and include only Planned Relative Time after Baseline.


Protocol : 204847
Population : Safety

Table 2.8

Summary of Haematology Values

Note to programmer: Please use the shell from Table 2.6.


Protocol : 204847
Population : Safety

Table 2.9

Summary of Haematology Change from Baseline

Note to programmer: Please use the shell from Table 2.6 and include only Planned Relative Time after Baseline.

Example : UR3 Page 1 of n

Protocol : 204847
Population : Safety

Table 2.10 Summary of Urinalysis Dipstick Results

Study Part: 1

| | Planned | | GSK3342830 250 mg | GSK3342830 500 mg | | Placebo |
|---|---|---|---|---|---|---|
| Test | Relative Time | Result | (N=xx) | (N=xx) | (N=xx) | (N=XX) |
| Urine General<br>Dipstick | Baseline | Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Negative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | No Result | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Not Done | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Day 2 | | ••• | • • • | • • • | |
| | Follow-up | • • • | ••• | ••• | • • • | • • • |
| Urine Occult<br>Blood<br>(Dipstick) | Baseline | None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Trace | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 1+ | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 2+ | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 3+ | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 4+ | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | 5+ | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | No Result | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Not Done | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

... ...

Note to Programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.

Example : EG1
Protocol : 204847
Population : Safety


Table 2.11 Summary of ECG Findings

Study Part: 1

| | GSK3342830 250 mg | GSK3342830 500 mg | | Total |
|---|---|---|---|---|
| | (N=XX) | (N=XX) | | (N=XX) |
| Baseline | | | | |
| n | XX | XX | | XX |
| Normal | xx (xx%) | xx (xx%) | | xx (xx%) |
| Abnormal, not clinically significant | xx (xx%) | xx (xx%) | ••• | xx (xx%) |
| Abnormal, clinically significant | xx (xx%) | xx (xx%) | • • • | xx (xx%) |
| Day 1 - 0.5 HR | | | | |
| n | XX | XX | | XX |
| Normal | xx (xx%) | xx (xx%) | | xx (xx%) |
| Abnormal, not clinically significant | xx (xx%) | xx (xx%) | ••• | xx (xx%) |
| Abnormal, clinically significant | xx (xx%) | xx (xx%) | | xx (xx%) |
| ••• | • • • | ••• | | ••• |

Note to Programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages. Timepoints for Part 1 and Part 3 are Baseline, Day 1-0.5 HR, Day 1-1 HR, Day 1-1.5 HR, Day 1-2 HR, Day 1-3 HR, Day 1-4 HR, Day 1-6 HR, Day 1-12 HR, Day 1-12 HR, Day 1-12 HR, Day 1-14 HR, Da

Note: Baseline is defined as the last nonmissing measurement before dosing.

Unscheduled measurements are not included in this summary table except when calculating baseline.

Example : EG2
Protocol : 204847
Population : Safety


Table 2.12 Summary of ECG Values

Study Part: 1

| ECG Test | Group | N | Planned Relative Time | n | Mean | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXXXX (XXX) | GSK3342830 250 mg | XXX | Baseline<br>Day 1 - 0.5 HR | xx<br>xx | XX.X<br>XX.X | xx.xx<br>xx.xx | xx<br>xx | xx<br>xx | XX<br>XX |
| | | | Follow-Up | XX | XX.X | XX.XX | xx | XX | XX |
| XXXXXXXX (XXX) | GSK3342830 500 mg | XXX | Baseline | XX | XX.X | XX.XX | XX | XX | XX |
| XXXXXXXX (XXX) | | XXX | Baseline | xx | xx.x | xx.xx | XX | xx | XX |

Note to Programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages. Timepoints for Part 1 and Part 3 are Baseline, Day 1-0.5 HR, Day 1-1 HR, Day 1-1.5 HR, Day 1-2 HR, Day 1-3 HR, Day 1-4 HR, Day 1-6 HR, Day 1-1.5

Note: Baseline is defined as the last nonmissing measurement before dosing for the respective treatment period Unscheduled measurements are not included in this summary table except when calculating baseline.

Example : EG2 Page 1 of n

Protocol : 204847
Population : Safety

Table 2.13
Summary of Change from Baseline in ECG Values

Note to programmer: Please use the shell from Table 2.12 and include only Planned Relative Time after Baseline.

Example : SAFE\_T1
Protocol : 204847
Population : Safety


Table 2.14
Summary of Frequency of Maximum Post-Dose ECG Parameter Corrected QTc Interval

Study Part: 1

| | GSK3342830 250 mg<br>(N=XX) | GSK3342830 550 mg<br>(N=XX) | <br>(N=XX) | Placebo<br>(N=XX) |
|---|---|---|---|---|
| QTcB (msec) | | | | |
| n | XX | XX | xx | XX |
| <=450 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >450-<=479 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >=480-<=499 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >=500 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| QTcF (msec) | | | | |
| n | XX | XX | xx | XX |
| <=450 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >450-<=479 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >=480-<=499 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >=500 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note to Programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.

Example : SAFE\_T1 Page 1 of n

Protocol : 204847
Population : Safety

Table 2.15
Summary of Frequency of Maximum Change from Baseline for ECG Parameter Corrected QTc Interval

Study Part: 1

| | GSK3342830 250 mg | GSK3342830 550 mg | | Placebo |
|-------------|-------------------|-------------------|----------|----------|
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| QTcB (msec) | | | | |
| n | XX | XX | XX | XX |
| <=30 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >30-<=59 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >=60 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| QTcF (msec) | | | | |
| n | XX | XX | XX | XX |
| <=30 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >30-<=59 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >=60 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note to Programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages.

Note: Baseline is defined as the last nonmissing measurement before dosing for the respective treatment period.

Unscheduled measurements are not included in this summary table except when calculating baseline.

Example : VS1
Protocol : 204847
Population : Safety


Table 2.16
Summary of Vital Signs

Study Part: 1

| Vital Sign | Group | N | Planned Relative Time | n | Mean | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXXXX (XXX) | GSK3342830 250 mg | XXX | Baseline<br>Day 1 - 0.5 HR | XX<br>XX | XX.X<br>XX.X | XX.XX<br>XX.XX | XX<br>XX | XX<br>XX | XX<br>XX |
| | | | <br>Follow-Up | XX | XX.X | XX.XX | xx | XX | XX |
| XXXXXXXX (XXX) | GSK3342830 500 mg | XXX | Baseline | xx | xx.x | xx.xx | xx | xx | XX |
| XXXXXXXX (XXX) | | XXX | Baseline | xx | xx.x | xx.xx | xx | xx | xx |

Note to Programmer: Continue for all treatments in Part 1, Part 2, and Part 3. Present Part 2 and Part 3 on separate pages. Timepoints for Part 1 and Part 3 are Baseline, Day 1-0.5 HR, Day 1-1 HR, Day 1-1.5 HR, Day 1-2 HR, Day 1-3 HR, Day 1-4 HR, Day 1-6 HR, Day 1-12 HR, Day 1-12 HR, Day 1-12 HR, Day 1-12 HR, Day 1-14 HR, Da

Note: Baseline is defined as the last nonmissing measurement before dosing.

Unscheduled measurements are not included in this summary table except when calculating baseline.


Protocol : 204847
Population : Safety

Table 2.17

Summary of Change from Baseline in Vital Signs

Note to programmer: Please use the shell from Table 2.14 and include only Planned Relative Time after Baseline.

: PK01 Example Page 1 of n Protocol : 204847

Population : PK

Table 3.01 Summary of GSK3342830 Single Dose Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment in Part 1 and Part 3

Part: Part 1

| | Study Day | | Planned<br>Relative | | No. | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose | | N | Time | n | Imputed | Mean | SD | CV% | Median | Min. | Max. |
| xxx mg | 1 | XX | pre-dose | XX | XX | NQ | • | • | • | | • |
| | | | 0.5h | XX | 0 | xxxx.x | XX.XX | XX.X | XXXX.X | XXXX | XXXX |
| | | | 1h | XX | 0 | XXXX.X | XX.XX | XX.X | XXXX.X | XXXX | XXXX |
| | | | 1.25h | XX | 0 | XXXX.X | XX.XX | XX.X | XXXX.X | XXXX | XXXX |
| | | | 1.5h | XX | 0 | XXXX.X | XX.XX | XX.X | XXXX.X | XXXX | XXXX |

point and 0.5, 1,1.25,1.5, 2, 2.5, 3,3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24,36 and 48 hours after dosing. If mean is below the level of quantification, report the mean value as NQ.

Example : PK01 Protocol : 204847

Population : PK

Table 3.02
Summary of GSK3342830 Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment in Part 2


| Dose | Day | N | Planned<br>Relative<br>Time | n | No.<br>Imputed | Mean | SD | CV% | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx mg | 1 | XX | pre-dose | XX | XX | NQ | • | - | • | • | |
| | | | 0.5h | XX | 0 | XXXX.X | XX.XX | XX.X | XXXX.X | XXXX | XXXX |
| | | | 1h | XX | 0 | XXXX.X | XX.XX | XX.X | XXXX.X | XXXX | XXXX |
| | | | 1.25h | XX | 0 | xxxx.x | XX.XX | XX.X | XXXX.X | XXXX | XXXX |
| | | | 1.5h | XX | 0 | XXXX.X | XX.XX | xx.x | xxxx.x | XXXX | XXXX |
| | | | ••• | | | | | ••• | | | |
| | 15 | XX | pre-dose | XX | XX | NQ | | • | • | • | • |
| | | | 0.25h | XX | 0 | XXXX.X | XX.XX | xx.x | xxxx.x | XXXX | xxxx |
| | | | ••• | | | | ••• | | | | |

Note to Programmer: Blood samples for PK analysis on day 1 will be collected at predose, 0.5, 1.25,1.5, 2,2.5,3,3.5,4,4.5,5,6,8,10,12,16 and 24. Timepoints on day 15 is Pre-dose,0.5,1,1.25,1.5,2,2.5,3,3.5,4,4.5, 5,6 and 8.If mean is below the level of quantification, report the mean value as NQ.


Protocol : 204847
Population : PK Parameter

Table 3.03

 $\hbox{Summary of Untransformed GSK3342830 Single Dose Plasma Pharmacokinetic Parameters in Part 1 and Part 3 } \\$ 

#### Part: Part 1

| | Summary | | | Dose 1 | evel | | |
|---|---|---|---|---|---|---|---|
| Parameter | Statistics | XX mg | XX mg | XX mg | XX mg | XX mg | XX mg |
| Cmax (units) | N | xx | XX | XX | XX | XX | XX |
| | n | xx | XX | XX | XX | XX | XX |
| | Arithmetic Mean | xxxx.xx | xxxx.xx | xxxx.xx | XXXX.XX | XXXX.XX | xxxx.xx |
| | 95% CI | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) |
| | SD | xxxx.xxx | xxxx.xxx | xxxx.xxx | XXXX.XXX | XXXX.XXX | xxxx.xxx |
| | Median | xxxx.xx | xxxx.xx | xxxx.xx | XXXX.XX | XXXX.XX | xxxx.xx |
| | Min | xxx | XXX | XXX | XXX | XXX | xxx |
| | Max | xxx | XXX | XXX | XXX | XXX | xxx |

Note to Programmer: Present all Part 1 first, then repeat for Part 3 Additional untransformed parameters include AUC(0-t), AUC(0- $\infty$ ), Tmax, t1/2, CL, Vss, %AUCex, tlast, lambda\_z, lambda\_z\_lower, lambda\_z\_upper, lambda\_z\_no. of points.

Protocol : 204847

Population : PK Parameter

Table 3.04

Summary of Log-transformed GSK3342830 Single Dose Plasma Pharmacokinetic Parameters in Part 1 and Part 3

# Part: Part 1

| | Summary | | Dose level | | | | |
|---|---|---|---|---|---|---|---|
| Parameter | Statistics | XX mg | XX mg | XX mg | XX mg | XX mg | XX mg |
| Cmax (units) | N | XX | XX | XX | XX | XX | XX |
| | n | XX | XX | xx | XX | XX | XX |
| | Geometric Mean | xxxx.xx | xxxx.xx | xxxx.xx | XXXX.XX | XXXX.XX | XXXX.XX |
| | 95% CI | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) |
| | Geometric SD | xxxx.xxx | xxxx.xxx | xxxx.xxx | XXXX.XXX | XXXX.XXX | XXXX.XXX |
| | %CVb | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx |

Note to Programmer: Present all Part 1 first, then repeat for Part 3 Additional untransformed parameters include AUC(0-t), AUC(0- $\infty$ ), t1/2, CL, Vss.

Protocol : 204847

Population : PK Parameter

Table 3.05
Summary of Untransformed GSK3342830 Single Dose Urine Pharmacokinetic Parameters in Part 1 and Part 3

Part: Part 1

| | Summary | | Dose level | | | | |
|---|---|---|---|---|---|---|---|
| Parameter | Statistics | XX mg | XX mg | XX mg | XX mg | XX mg | XX mg |
| Ae (units) | N | XX | XX | XX | XX | XX | XX |
| | n | XX | XX | XX | XX | XX | XX |
| | Geometric Mean | xxxx.xx | xxxx.xx | xxxx.xx | XXXX.XX | XXXX.XX | XXXX.XX |
| | 95% CI | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) |
| | Geometric SD | xxxx.xxx | xxxx.xxx | xxxx.xxx | XXXX.XXX | XXXX.XXX | XXXX.XXX |
| | %CVb | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx | xxxx.xx |

Note to Programmer: Present all Part 1 first, then repeat for Part 3 Additional untransformed parameters include Clr, Feu(0-4) (units), Feu(4-8) (units), Feu(8-12) (units), Feu(12-24) (units), Feu(24-48) (units).

Example : PKPT1 Protocol : 204847

Population : PK Parameter

 ${\tt Table~3.06}\\ {\tt Summary~of~Untransformed~GSK3342830~Plasma~Pharmacokinetic~Parameters~in~Part~2}\\$ 


| | | Summary | | | Dose 1 | evel | | |
|---|---|---|---|---|---|---|---|---|
| Day | Parameter | Statistics | XX mg | XX mg | XX mg | XX mg | XX mg | XX mg |
| 1 | | | | | | | | |
| 1 | Cmax (units) | N | XX | XX | XX | XX | XX | XX |
| | | n | XX | XX | XX | XX | XX | XX |
| | | Arithmetic | xxxx.xx | XXXX.XX | xxxx.xx | XXXX.XX | XXXX.XX | XXXX.XX |
| | | Mean | | | | | | |
| | | 95% CI | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) |
| | | SD | XXXX.XXX | XXXX.XXX | XXXX.XXX | XXXX.XXX | XXXX.XXX | XXXX.XXX |
| | | Median | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | | Min | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Max | XXX | XXX | XXX | XXX | XXX | XXX |

### Note to Programmer:

Additional untransformed parameters include AUC(0-t), AUC(0- $\infty$ ), AUC(0- $\tau$ ), Tmax, t1/2, CL, Vss, %AUCex, tlast, lambda\_z, lambda z lower, lambda z upper, lambda z no. of points, C $\tau$ , Ratio of time invariance, Ratio of accumulation. Repeat for day 15

Example : PKPT3
Protocol : 204847

Population : PK Parameter


Table 3.07
Summary of Log-transformed GSK3342830 Plasma Pharmacokinetic Parameters in Part 2

| | | Summary | | | Dose | Dose level | | |
|---|---|---|---|---|---|---|---|---|
| Day | Parameter | Statistics | XX mg | XX mg | XX mg | XX mg | XX mg | XX mg |
| 1 | <br>Cmax<br>(units) | N | xx | xx | xx | xx | xx | xx |
| | | n | XX | XX | XX | XX | XX | XX |
| | | Geometric Mean<br>95% CI | xxxx.xx<br>(xxxx.x,xxxx.x) | xxxx.xx<br>(xxxx.x,xxxx.x) | xxxx.xx<br>(xxxx.x,xxxx.x) | xxxx.xx<br>(xxxx.x,xxxx.x) | xxxx.xx<br>(xxxx.x,xxxx.x) | xxxx.xx<br>(xxxx.x,xxxx.x) |
| | | Geometric SD %CVb | xxxx.xxx<br>xxxx.xx | xxxx.xxx<br>xxxx.xx | xxxx.xxx<br>xxxx.xx | xxxx.xxx<br>xxxx.xx | xxxx.xxx<br>xxxx.xx | xxxx.xxx<br>xxxx.xx |

Note to Programmer:

Additional untransformed parameters include AUC(0-t), AUC(0- $\infty$ ), AUC(0- $\tau$ ), t1/2, CL, Vss, C $\tau$ . Repeat for Day 15.

Example : PKPT1

Protocol : 204847

Population : PK Parameter


| | | | Summary<br>Statistics | | | | |
|---|---|---|---|---|---|---|---|
| Day | Parameter | XX mg | XX mg | XX mg | XX mg | XX mg | XX mg |
| 1 | Ae (units) | XX | xx | XX | XX | XX | xx |
| | | XX | XX | XX | XX | XX | XX |
| | | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) | (xxxx.x, xxxx.x) |
| | | xxxx.xxx | xxxx.xxx | xxxx.xxx | XXXX.XXX | XXXX.XXX | XXXX.XXX |
| | | xxxx.xx | xxxx.xx | XXXX.XX | XXXX.XX | XXXX.XX | xxxx.xx |

Note to Programmer:

Additional untransformed parameters include Clr, Feu(0-8) (units), Feu(8-24) (units). Repeat for Day 15.

Protocol : 204847

Population : PK Parameter

Table 3.09
Summary of Statistical Analysis of GSK3342830 Plasma Dose Proportionality in Part 1

| Dose (units) | Parameter | Estimated Slope for log(dose) | Standard<br>Error | 90% CI<br>Lower-Upper | P-Value<br>(b=1) |
|---|---|---|---|---|---|
| XX mg | Cmax<br>(units) | x.xxx | x.xxx | x.xxxx-x.xxxx | x.xxxx |
| | | x.xxx | x.xxx | x.xxxx-x.xxxx | x.xxxx |

Note: The power model, log(parameter) = log(a) + b\*log(dose), was used to estimate the slope, corresponding 90% confidence interval, and the p-value testing dose proportionality (b=1). Natural log-transformation was used.

Source Data: Listing 44.

Note to programmer: In the case where dose proportionality is not established over the entire dosing range, secondary analysis of dose proportionality will be assessed for select doses over the higher dosing range with the power model or by pair-wise analysis of variance (ANOVA) using the SAS mixed models procedure. If the secondary analysis using the pair-wise ANOVA approach is performed, a reference dose would be chosen based on the lowest clinically relevant dose over which the pharmacokinetics can be adequately described and the other doses would be treated as test doses.

Protocol : 204847

Population : PK Parameter

\_

| Day | Dose<br>(Units) | Parameter | Estimated Slope for log(dose) | Standard<br>Error | 90% CI<br>Lower-Upper | P-Value<br>(b=1) |
|---|---|---|---|---|---|---|
| 15 | XX mg | Cmax<br>(units) | x.xxx | x.xxx | x.xxxx-x.xxxx | x.xxx |
| | | | X.XXX | X.XXX | x.xxxx-x.xxxx | x.xxxx |

Note: The power model, log(parameter) = log(a) + b\*log(dose), was used to estimate the slope, corresponding 90% confidence interval, and the p-value testing dose proportionality (b=1). Natural log-transformation was used.

Source Data: Listing 46.

Note to programmer: In the case where dose proportionality is not established over the entire dosing range, secondary analysis of dose proportionality will be assessed for select doses over the higher dosing range with the power model or by pair-wise analysis of variance (ANOVA) using the SAS mixed models procedure. If the secondary analysis using the pair-wise ANOVA approach is performed, a reference dose would be chosen based on the lowest clinically relevant dose over which the pharmacokinetics can be adequately described and the other doses would be treated as test doses.

Example : PK\_T1
Protocol : 204847

Population : PK Parameter

Table 3.11
Summary of Statistical Analysis of GSK3342830 Plasma Time Invariance in Part 2


Dose: XX mg

| | | | | | Ratio of | 90% Confidence | |
|---|---|---|---|---|---|---|---|
| | | | Geometric | Regimen | Geometric | Interval of | |
| Parameter (Unit) | Day | N | LS Means | Comparison | LS Means (%) | Ratio (%) | CVw(%) |
| AUC(0-inf) (Unit) | 1 | XX | X.XXX | 15/1 | X.XXX | (x.xxx, x.xxx) | X.XXX |
| AUC(0-tau) (Unit) | 15 | XX | X.XXX | | | | |

# Notes to programmer: Repeat for each dose level.

Note: A linear mixed-effect model with group (group=1 for AUC(0-inf) on Day 1, and group=2 for AUC(0-tau) on Day 15) as a fixed effect and subject as a random effect was fitted to the natural log transformed PK parameters.

Source Data: Listing 46.

Example : PK T1 Page 1 of n

Protocol : 204847
Population : PK Parameter

 ${\tt Table 3.12}\\ {\tt Summary of Statistical Analysis of GSK3342830~Plasma~Accumulation~Ratio~in~Part~2}\\$ 

| Parameter<br>(Unit) | Dose*<br>(mg) | Day | N | Geometric<br>LS Means | Regimen<br>Comparison | Ratio of<br>Geometric<br>LS Means (%) | 90% Confidence<br>Interval of<br>Ratio (%) | CVw (%) |
|---|---|---|---|---|---|---|---|---|
| AUC(0-tau) (Unit) | XX | 1 | XX | x.xxx | 15/1 | x.xxx | (x.xxx, x.xxx) | x.xxx |
| | | 15 | XX | X.XXX | | | | |
| | УУ | 1 | XX | X.XXX | 15/1 | x.xxx | (x.xxx, x.xxx) | |
| | | 15 | XX | X.XXX | | | | |
| | ZZ | 1 | XX | X.XXX | 15/1 | X.XXX | (x.xxx, x.xxx) | |
| | | 15 | XX | X.XXX | | | | |

Note: A linear mixed-effect model with dose, day, and dose-by-day interaction as fixed effects and subject as a random effect was fitted to the natural log transformed PK parameters.

Source Data: Listing 46.

<sup>\*</sup> If dose-by-day interaction is significant (p-value less then 0.05), then point estimate and 90% CI will be reported for each dose level.

Example : PK T1 Protocol : 204847

Population : PK Parameter

Table 3.13 Summary of Statistical Analysis of GSK3342830 Plasma Steady State Assessment in Part 2

| | | Estimated Slope | 90% CI |
|-----------------|---------------------|-----------------|---------------|
| Parameter | Days Included | for Day | Lower-Upper |
| Ctrough (units) | 3, 6, 9, 12, 13, 15 | X.XXX | x.xxxx-x.xxxx |


Note to programmer: If the 90% CI does not include zero, repeat the analysis without the data for the earliest day used in the previous analysis. Display the results for all models run.

Note: A mixed effect model will be fitted by dose and day (as a continuous covariate) as a fixed effect term and subject as a random effect term. No formal statistical hypothesis tested. Steady state is estimated to be achieved by the earliest day included in the analysis when the 90% CI of the slope includes 0.

Source Data: Table 3.06.

Example : PK\_T2
Protocol : 204847

Population : PK Parameter

| PK Parameter on log scale<br>Model Parameter | Mean | SD | MC error | 5 <sup>th</sup> Percentile | Median | 95 <sup>th</sup> Percentile |
|---|---|---|---|---|---|---|
| AUC[0-t](µg.h/mL) | | | | | | |
| Intercept | XXXX.X | XXXX.X | XXXX.X | XXXX.X | xxxx.x | XXXX.X |
| Slope of log dose | XXXX.X | xxxx.x | xxxx.x | xxxx.x | XXXX.X | xxxx.x |
| Precision | XXXX.X | xxxx.x | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| Cmax (µg/mL) | | | | | | |
| Intercept | XXXX.X | xxxx.x | xxxx.x | xxxx.x | XXXX.X | XXXX.X |
| Slope of log dose | XXXX.X | xxxx.x | xxxx.x | xxxx.x | XXXX.X | XXXX.X |
| Precision | XXXX.X | xxxx.x | XXXX.X | xxxx.x | XXXX.X | XXXX.X |


Note: The posterior distributions are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term.

Programmer note: Decimals will be adjusted to include approximately 5 significant digits.

Example : PK\_T2
Protocol : 204847

Population : PK Parameter

| PK Parameter on log scale<br>Model Parameter | Mean | SD | MC error | 5 <sup>th</sup> Percentile | Median | 95 <sup>th</sup> Percentile |
|---|---|---|---|---|---|---|
| AUC[0-8]x3(μg.h/mL) | | | | | | |
| Intercept | XXXX.X | xxxx.x | xxxx.x | xxxx.x | XXXX.X | xxxx.x |
| Slope of log dose | XXXX.X | xxxx.x | xxxx.x | XXXX.X | XXXX.X | xxxx.x |
| Precision | XXXX.X | XXXX.X | XXXX.X | xxxx.x | XXXX.X | XXXX.X |
| Cmax (µg/mL) | | | | | | |
| Intercept | XXXX.X | xxxx.x | xxxx.x | xxxx.x | XXXX.X | xxxx.x |
| Slope of log dose | XXXX.X | XXXX.X | xxxx.x | xxxx.x | XXXX.X | xxxx.x |
| Precision | XXXX.X | xxxx.x | xxxx.x | xxxx.x | XXXX.X | XXXX.X |


Note: The posterior distributions are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term.

Programmer note: Decimals will be adjusted to include approximately 5 significant digits.

Example : PK\_T3
Protocol : 204847

Population : PK Parameter

Table 3.16
Summary of PK Parameters for Part 1 - Bayesian Prediction of Individual Subjects


| PK Parameter | 250 mg | 500 mg | 1000 mg | 2000 mg | 4000 mg | 6000 mg |
|---|---|---|---|---|---|---|
| Statistics | | | | | | |
| AUC[0-t] (µg.h/mL) | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | XXX |
| Observed Mean | XXXX.X | XXXX.X | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| Predictive Distributi | on | | | | | |
| Mean | XXXX.X | XXXX.X | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| 5 <sup>th</sup> Percentile | XXXX.X | xxxx.x | xxxx.x | xxxx.x | xxxx.x | XXXX.X |
| Median | XXXX.X | xxxx.x | xxxx.x | xxxx.x | xxxx.x | XXXX.X |
| 95 <sup>th</sup> Percentile | xxxx.x | XXXX.X | XXXX.X | XXXX.X | XXXX.X | xxxx.x |
| Cmax (µg/mL) | | | | | | |
| Observed Mean | XXXX.X | xxxx.x | xxxx.x | xxxx.x | xxxx.x | XXXX.X |
| Predictive Distributi | on | | | | | |
| Mean | XXXX.X | xxxx.x | xxxx.x | xxxx.x | xxxx.x | XXXX.X |
| 5 <sup>th</sup> Percentile | XXXX.X | xxxx.x | xxxx.x | xxxx.x | xxxx.x | XXXX.X |
| Median | XXXX.X | xxxx.x | xxxx.x | xxxx.x | xxxx.x | XXXX.X |
| 95 <sup>th</sup> Percentile | xxxx.x | xxxx.x | xxxx.x | xxxx.x | xxxx.x | XXXX.X |

Note: The predictive distributions are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term.

### Programming notes:

- 1. Decimals will be adjusted to include approximately 5 significant digits as a guideline not as a requirement.
- 2. If no observed values available for some doses, use 'NA' for the observed mean/n.

Example :  $PK_T4$  Page 1 of n Protocol :  $20\overline{4}847$ 

Population : PK Parameter

Table 3.17
Summary of PK Parameters for Part 2 - Bayesian Prediction of Individual Subject

| PK Parameter | 1000 mg | 2000 mg | 4000 mg |
|-----------------------------|---------|---------|---------|
| Statistics | - | - | - |
| AUC[0-8]x3 (µg.h/mL) | | | |
| n | XXX | XXX | xxx |
| Observed Mean | XXXX.X | XXXX.X | XXXX.X |
| Predictive Distribution | | | |
| Mean | XXXX.X | xxxx.x | xxxx.x |
| 5 <sup>th</sup> Percentile | XXXX.X | XXXX.X | xxxx.x |
| Median | XXXX.X | XXXX.X | xxxx.x |
| 95 <sup>th</sup> Percentile | XXXX.X | XXXX.X | xxxx.x |
| Cmax (µg/mL) | | | |
| Observed Mean | XXXX.X | XXXX.X | XXXX.X |
| Predictive Distribution | | | |
| Mean | xxxx.x | xxxx.x | XXXX.X |
| 5 <sup>th</sup> Percentile | xxxx.x | xxxx.x | XXXX.X |
| Median | xxxx.x | xxxx.x | XXXX.X |
| 95 <sup>th</sup> Percentile | XXXX.X | XXXX.X | XXXX.X |

Note: The predictive distributions are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term.

Programming notes: Decimals will be adjusted to include approximately 5 significant digits.

Example : PK\_T4
Protocol : 204847

Population : PK Parameter

Table 3.18
Summary of PK Parameters for Part 1 - Bayesian Predictive Probability

| PK Parameter | Threshold on actual scale | | Probab | Probability (greater than threshold | | | |
|---|---|---|---|---|---|---|---|
| | | 250 mg | 500 mg | 1000 mg | 2000 mg | 4000 mg | 6000 mg |
| AUC[0-t] (µg.h/mL) | 3460 | x.xx% | X.XX% | X.XX% | X.XX% | xx.xx% | xx.xx% |
| Cmax (µg/mL) | 2590 | x.xx% | x.xx% | x. xx% | X.XX% | xx.xx% | xx.xx% |


Note: The predictive distributions are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term.

Note: Each probability is the posterior predictive probability of the PK parameter exceeding the threshold, for a hypothetical future study subject.

#### Programming notes:

Example : PK\_T4
Protocol : 204847

Population : PK Parameter

Table 3.19
Summary of PK Parameters for Part 2 - Bayesian Predictive Probability

| PK Parameter | Threshold on actual scale | eater than threshold ob | served data) | |
|---|---|---|---|---|
| | 56426 | 1000 mg | 2000 mg | 4000 mg |
| AUC[0-8]x3 (µg.h/mL) | 3460 | x.xx% | x.xx% | xx.xx% |
| Cmax (µg/mL) | 2590 | x.xx% | X.XX% | xx.xx% |


Note: The predictive distributions are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term.

Note: Each probability is the posterior predictive probability of the PK parameter exceeding the threshold, for a hypothetical future study subject.

### Programming notes:


Protocol : 204847
Population : PK Parameter

| PK Parameter | Threshold on actual scale | | Probability (greater than threshold observed data) | | | | |
|---|---|---|---|---|---|---|---|
| | | 250 mg | 500 mg | 1000 mg | 2000 mg | 4000 mg | 6000 mg |
| AUC[0-t] (µg.h/mL) | 2875 | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |
| Cmax (µg/mL) | 2270 | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |

Note: The inferential probability are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term.

Note: Each probability is the posterior inferential probability of the mean PK parameter exceeding the threshold.

### Programming notes:


Protocol : 204847
Population : PK Parameter

Table 3.21

Summary of PK Parameters for Part 2 - Bayesian Inferential Probability

Protocol : 204847

| PK Parameter | Threshold on actual scale | Probability (greater than threshold observed data) | | |
|---|---|---|---|---|
| | | 1000 mg | 2000 mg | 4000 mg |
| AUC[0-8]x3 (µg.h/mL) | 2875 | 0.xxxx | 0.xxxx | 0.xxxx |
| Cmax (µg/mL) | 2270 | 0.xxxx | 0.xxxx | 0.xxxx |

Note: The inferential distributions are derived from linear model log-PK-parameter = intercept + slope\*log-dose + error term.

Note: Each probability is the posterior inferential probability of the mean PK parameter exceeding the threshold.

### Programming notes:

Protocol : 204847

Population : PK Parameter

Table 3.22 Summary of Statistical Analysis of GSK3342830 Single Dose Plasma Pharmacokinetic Parameters in Part 1 and Part 3 Subjects

| Parameter (Unit) | Dose<br>(mg) | Study Part | N | Geometric<br>LS Means | Regimen<br>Comparison | Ratio of<br>Geometric<br>LS Means (%) | 90% Confidence<br>Interval of<br>Ratio (%) |
|---|---|---|---|---|---|---|---|
| AUC(0-t)<br>(Unit) | XX | Part 1 | XX | X.XXX | Part 3/Part 1 | x.xxx | (x.xxx, x.xxx) |
| AUC(0-inf)<br>(Unit) | УУ | Part 3<br>Part 1 | XX | x.xxx<br>x.xxx | Part 3/Part 1 | x.xxx | (x.xxx, x.xxx) |
| Cmax (Unit) | ZZ | Part 3<br>Part 1<br>Part 3 | XX<br>XX<br>XX | x.xxx<br>x.xxx<br>x.xxx | Part 3/Part 1 | x.xxx | (x.xxx, x.xxx) |

Note: A linear mixed-effect model with study part as fixed effect was fitted to the natural log transformed PK parameters.

Part 1 subjects were normal healthy volunteers and Part 3 subjects were Japanese healthy volunteers.

Source Data: Listing 44.